CLINICAL TRIAL: NCT01557244
Title: A 24-WEEK RANDOMIZED, OPEN-LABEL, STUDY TO EVALUATE THE SAFETY AND EFFICACY OF FESOTERODINE IN SUBJECTS AGED 6 TO 17 YEARS WITH SYMPTOMS OF DETRUSOR OVERACTIVITY ASSOCIATED WITH A NEUROLOGICAL CONDITION (NEUROGENIC DETRUSOR OVERACTIVITY)
Brief Title: A Study To Find Out How Fesoterodine Works In Children Aged 6 To 17 Years With Bladder Overactivity Caused By A Neurological Condition
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A0221047; 2010-022475-55 (EudraCT Number)
Record Dates: First submitted 2012-03-15; First posted 2012-03-19 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2020-12

CONDITIONS: Urinary Bladder, Neurogenic
Keywords: neurogenic detrusor overactivity; neurogenic bladder; neuropathic bladder; neurologic disease; fesoterodine
MeSH Terms: conditions — Urinary Bladder, Neurogenic | interventions — oxybutynin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Fesoterodine PR 4 mg (Experimental): Fesoterodine PR 4 mg for 12 weeks in active comparator period, followed by 12 weeks in safety extension period
  Interventions: Drug: Fesoterodine PR 4 mg
- Fesoterodine PR 8 mg (Experimental): Fesoterodine 8 mg for first week followed by 11 weeks at 8 mg in active control period, followed by 12 weeks in safety extension period.
  Interventions: Drug: Fesoterodine PR 8 mg
- Oxybutynin (Active Comparator): Oxybutynin
  Interventions: Drug: Oxybutynin; Drug: Fesoterodine PR
- Fesoterodine BIC 2 mg (Experimental): Fesoterodine BIC 2 mg for 12 weeks in efficicay period, followed by 12 weeks in safety extension period.
  Interventions: Drug: Fesoterodine BIC 2 mg
- Fesoterodine BIC 4 mg (Experimental): Fesoterodine BIC 4 mg for first week followed by 11 weeks at 8 mg in the efficacy period, followed by 12 weeks in safety extension period.
  Interventions: Drug: Fesoterodine BIC 4 mg

INTERVENTIONS:
Drug: Fesoterodine PR 4 mg — Fesoterodine 4 mg tablet once daily for 24 weeks
  Arms: Fesoterodine PR 4 mg
Drug: Fesoterodine PR 8 mg — Fesoterodine PR 8 mg tablet once daily for 24 weeks, the first week being 4 mg.
  Arms: Fesoterodine PR 8 mg
Drug: Fesoterodine PR 8 mg — Fesoterodine 8 mg tablet once daily for 24 weeks, the first week being 4 mg.
  Arms: Fesoterodine PR 8 mg
Drug: Oxybutynin — Oxybutynin extended release tablets according to approved pediatric labeling for 12 weeks with dose titration phase for first 4 weeks to achieve dose optimisation.
  Arms: Oxybutynin
Drug: Fesoterodine PR — Fesoterodine 4 mg or 8 mg tablets once daily for 12 weeks after 12 weeks of oxybutinin. Those assigned to 8 mg will take 4 mg for the first week.
  Other Names: Safety extension phase
  Arms: Oxybutynin
Drug: Fesoterodine BIC 2 mg — Fesoterodine BIC 2 mg tablet once daily for 24 weeks.
  Arms: Fesoterodine BIC 2 mg
Drug: Fesoterodine BIC 4 mg — Fesoterodine BIC 4 mg tablet once daily for 24 weeks, with the first week being 2 mg.
  Arms: Fesoterodine BIC 4 mg

SUMMARY:
The objective of the study is to find out if the medicine fesoterodine is a useful treatment in children with bladder muscle overactivity caused by a neurological condition. Children will be aged 6 to 17 years old. This is done by finding out how well it works, what the body does to fesoterodine, what side effects are experienced and the safety of fesoterodine. It will be compared with the medicine oxybutynin, which is already available for treating the condition.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 6 to 17 years old
* Subjects with stable neurological disease and neurogenic detrusor overactivity
* Subjects using clean intermittent catheterization may participate

Exclusion Criteria:

* Concomitant medications which may increase the risk to subjects or confound study results
* Other medical conditions which may increase the risk to subjects or confound study results
* Contraindications to the use of fesoterodine or oxybutynin

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 181 (Actual)
Dates: Start 2012-07-02 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2020-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (84):
- United States (18):
  - Urological Associates of Southern Arizona, Tucson, Arizona
  - Childrens Hospital of Orange County, Orange, California
  - CHOC Children's Urology Center, Orange, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Georgia Urology, P.A., Atlanta, Georgia
  - Judson L. Hawk Jr. M.D., Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Loyola University Outpatient Center, Maywood, Illinois
  - The Iowa Clinic, West Des Moines, Iowa
  - UNC Chapel Hill Memorial Hospital, Chapel Hill, North Carolina
  - UNC Memorial Hospital Pediatric Clinic, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Liberty Township, Ohio
  - Advanced Radiology, East Providence, Rhode Island
  - Pharma Resource, East Providence, Rhode Island
  - University Urological Associates, Inc, Providence, Rhode Island
  - University Urological Associates, Inc., Providence, Rhode Island
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen, Urologie, Edegem, Antwerpen
  - Hôpital Universitaire des Enfants Reine Fabiola, Brussels, Brussels Capital
- Centre hospitalier universitaire (CHU) Sainte-Justine, Montreal, Quebec, Canada
- Tallinn Children's Hospital, Tallinn, Estonia
- Tampere University Hospital, Tampere, Finland
- France (3):
  - Centre d'Investigation Clinique, Bron
  - Groupement Hospitalier Est - Hopital Femme Mere Enfant, Bron
  - Hôpitaux Pédiatriques de Nice CHU-Lenval, Nice
- Kliniken Maria Hilf GmbH, Mönchengladbach, North Rhine-Westphalia, Germany
- Greece (2):
  - University General Hospital of Larisa/ Urology Department, Larissa
  - Aristotle University of Thessaloniki, Thessaloniki
- Department of Pediatrics, Christian Medical College and Hospital, Ludhiana, Punjab, India
- Italy (5):
  - I.R.C.C.S. - Ospedale "Casa Sollievo della Sofferenza" - Dipartimento Scienze Chirurgiche, San Giovanni Rotondo, Foggia
  - Azienda Ospedaliera G. Brotzu, Dipartimento di Medicina interna-, Cagliari
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - IRCCS Ospedale Pediatrico Bambino Gesù, Roma
  - ULSS 6 VICENZA - Ospedale San Bortolo di Vicenza, Vicenza
- Japan (13):
  - Aichi Children's Health and Medical Center, Ōbu, Aichi-ken
  - Chiba Children's Hospital, Chiba, Chiba, Japan
  - Fukuoka Children's Hospital, Fukuoka, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo prefectural Kobe Children's Hospital, Kobe, Hyōgo
  - Kanagawa Children's Medical Center, Yokohama, Kanagawa
  - Shinshu University Hospital, Matsumoto, Nagano
  - Osaka Medical Center and Research Institute for Maternal and Child Health, Izumi-shi, Osaka
  - Dokkyo Medical University Koshigaya Hospital, Koshigaya, Saitama
  - Shizuoka Children's Hospital, Shizuoka, Shizuoka
  - Dokkyo Medical University Hospital / Urology, Shimotsuga-gun, Tochigi
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - The University of Tokyo Hospital / Urology, Bunkyo-ku, Tokyo
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas klinikos, Kaunas
  - Children's Hospital, Affiliate of Vilnius University Hospital Santaros Klinikos, Vilnius
- Malaysia (2):
  - Hospital Selayang, Batu Caves, Selangor
  - Hospital Kuala Lumpur, Kuala Lumpur
- Philippine Children's Medical Center, Quezon City, NCR, Philippines
- Poland (2):
  - Klinika Chorob Nerek i Nadcisnienia Dzieci i Mlodziezy, Gdansk
  - Specjalistyczny Gabinet Lekarski Paweł Kroll, Poznan
- Russia (5):
  - FGBNU Scientific center of children health, Moscow, Russian Federation
  - Kazan State Medical University, Kazan', Tatarstan Republic
  - Children's Republican Clinical Hospital, Department of Pediatric Surgery, Kazan'
  - Scientific Research Institute of Urology named after N.A.Lopatkin of the Hertsen Federal Medical, Moscow
  - SSS - Research Clinical Institute of Pediatrics n.a. Academician Y.E.Veltishchev GBOU VPO, Moscow
- Slovakia (2):
  - J. BREZA MEDICAL s.r.o., Bratislava
  - Narodny ustav detskych chorob, Bratislava
- Red Cross Children's Hospital, Cape Town, Western Cape, South Africa
- South Korea (6):
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Korea University Guro Hospital, Seoul, Korea
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - ASAN Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (5):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Infantil Universitario Niño Jesus, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Universitari i Politecnic La Fe, Valencia
- Akademiska barnsjukhuset, Uppsala, Sweden
- Universitäts-Kinderspital beider Basel, Basel, Switzerland
- National Cheng Kung University Hospital, Tainan, Taiwan
- Turkey (Türkiye) (4):
  - Necmettin Erbakan Universitesi Meram Tip Fakultesi, Konya, Konya / Turkey
  - Ankara Universitesi Tip Fakultesi Ibni Sina Hastanesi, Ankara
  - Hacettepe Universitesi Tip Fakultesi Uroloji Anabilim Dali, Ankara
  - Istanbul Universitesi Istanbul Tip Fakultesi, Istanbul
- United Kingdom (3):
  - Leicester Royal Infirmary, Leicester
  - Alder Hey Children's Hospital, Liverpool
  - Sheffield Children's NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Sano Y, Shoji S, Shahin M, Sweeney K, Darekar A, Malhotra BK. Population Pharmacokinetic and Pharmacodynamic Modeling of Fesoterodine in Pediatric Patients with Neurogenic Detrusor Overactivity. Eur J Drug Metab Pharmacokinet. 2023 May;48(3):257-269. doi: 10.1007/s13318-023-00818-8. Epub 2023 Mar 9. PMID 36892754
- [Derived] Kitta T, Darekar A, Malhotra B, Shahin MH, Jones P, Lindsay M, Mallen S, Nieto A, Crook TJ. Fesoterodine treatment of pediatric patients with neurogenic detrusor overactivity: A 24-week, randomized, open-label, phase 3 study. J Pediatr Urol. 2023 Apr;19(2):175.e1-175.e10. doi: 10.1016/j.jpurol.2022.11.020. Epub 2022 Nov 29. PMID 36504158
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221047&StudyName=A%20Study%20To%20Find%20Out%20How%20Fesoterodine%20Works%20In%20Children%20Aged%206%20To%2017%20Years%20With%20Bladder%20Overactivity%20Caused%20By%20A%20Neurological%20Condi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study had 2 cohorts: cohort 1 had participants with body weight greater than (>) 25 kilogram (kg) and cohort 2 had participants with body weight less than or equal to (<=) 25 kg. There were 2 phases in each cohort: cohort 1- active comparator phase followed by safety extension phase; cohort 2- efficacy phase followed by safety extension phase.
Groups:
- Cohort 1: Fesoterodine 4 mg: Participants with body weight >25 kg were randomized to receive fesoterodine 4 milligram (mg) prolonged release (PR) tablet orally once daily for 12 weeks in active comparator phase. Active comparator phase was followed by safety extension phase, where participants continued to receive fesoterodine 4 mg PR tablet orally once daily for another 12 weeks.
- Cohort 1: Fesoterodine 4 mg Then 8 mg: Participants with body weight >25 kg were randomized to receive fesoterodine 4 mg PR tablet orally once daily for first 1 week and if this dose was tolerated well, participants received fesoterodine 8 mg PR tablet orally once daily for next 11 weeks in active comparator phase and if dose was not tolerated then participants were withdrawn from the study. Active comparator phase was followed by safety extension phase, where participants continued to receive fesoterodine 8 mg PR tablet orally once daily for another 12 weeks.
- Cohort 1: Oxybutynin: Participants with body weight >25 kg were randomized to receive oxybutynin extended release (ER) tablet, at a daily dose in accordance with approved pediatric labeling and accepted practice. Dose titration was done for first 4 weeks. After Week 4, participants remained on the optimized daily dose for next 8 weeks, in active comparator phase.
- Cohort 1: Oxybutynin Then Fesoterodine 4 mg: Participants with body weight >25 kg who were randomized to receive oxybutynin ER tablet, at a daily dose in accordance with approved pediatric labeling and accepted practice, in active comparator phase; were allocated by investigator to receive fesoterodine 4 mg PR tablet orally once daily for 12 weeks in the safety extension phase.
- Cohort 1: Oxybutynin Then Fesoterodine 4 mg Then 8 mg: Participants with body weight >25 kg who were randomized to receive oxybutynin ER tablet, at a daily dose in accordance with approved pediatric labeling and accepted practice, in active comparator phase; were allocated by investigator to receive fesoterodine 4 mg PR tablet orally once daily for first 1 week followed by fesoterodine 8 mg PR tablet orally once daily for another 11 weeks (if the fesoterodine 4 mg dose was well tolerated) in the safety extension phase and if dose was not tolerated then participants were withdrawn from the study.
- Cohort 2: Fesoterodine 2 mg: Participants with body weight <=25 kg were randomized to receive fesoterodine 2 mg beads-in-capsule (BIC) capsule orally once daily for 12 weeks in efficacy phase. Efficacy phase was followed by safety extension phase, where participants continued to receive fesoterodine 2 mg BIC capsules orally once daily for another 12 weeks.
- Cohort 2: Fesoterodine 2 mg Then 4 mg: Participants with body weight <=25 kg were randomized to receive fesoterodine 2 mg BIC capsule orally once daily for first 1 week and if this dose was tolerated well, participants received fesoterodine 4 mg BIC capsule orally once daily for next 11 weeks in efficacy phase and if dose was not tolerated then participants were withdrawn from the study. Efficacy phase was followed by safety extension phase, where participants continued to receive fesoterodine 4 mg BIC capsule orally once daily for another 12 weeks.
Period: Active Comparator/Efficacy Phase:12Weeks
Arm/Group | Cohort 1: Fesoterodine 4 mg | Cohort 1: Fesoterodine 4 mg Then 8 mg | Cohort 1: Oxybutynin | Cohort 1: Oxybutynin Then Fesoterodine 4 mg | Cohort 1: Oxybutynin Then Fesoterodine 4 mg Then 8 mg | Cohort 2: Fesoterodine 2 mg | Cohort 2: Fesoterodine 2 mg Then 4 mg
Started | 42 | 42 | 40 | 0 | 0 | 28 | 29
Treated | 42 | 42 | 40 | 0 | 0 | 28 | 29
Completed | 33 | 40 | 36 | 0 | 0 | 21 | 28
Not Completed | 9 | 2 | 4 | 0 | 0 | 7 | 1
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Protocol Violation | 2 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal By Parent/Guardian | 2 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Medication Error Without Associated AEs | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Insufficient Clinical Response | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Failure to Meet Randomization Criteria | 0 | 1 | 1 | 0 | 0 | 1 | 0
Not completed — Other | 2 | 0 | 2 | 0 | 0 | 0 | 0
Period: Safety Extension Phase: 12 Weeks
Arm/Group | Cohort 1: Fesoterodine 4 mg | Cohort 1: Fesoterodine 4 mg Then 8 mg | Cohort 1: Oxybutynin | Cohort 1: Oxybutynin Then Fesoterodine 4 mg | Cohort 1: Oxybutynin Then Fesoterodine 4 mg Then 8 mg | Cohort 2: Fesoterodine 2 mg | Cohort 2: Fesoterodine 2 mg Then 4 mg
Started | 33 | 40 | 0 (Did not receive oxybutynin in safety extension phase.) | 16 (Allocated from oxybutynin arm to this arm by investigator in safety extension phase.) | 20 (Allocated from oxybutynin arm to this arm by investigator in safety extension phase.) | 21 | 28
Treated | 30 | 37 | 0 | 16 | 20 | 20 | 28
Completed | 30 | 36 | 0 | 15 | 20 | 20 | 28
Not Completed | 3 | 4 | 0 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal By Parent/Guardian | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Medication Error Without Associated AEs | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Insufficient Clinical Response | 1 | 2 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all randomized participants.
Groups:
- Cohort 1: Fesoterodine 4 mg: Participants with body weight >25 kg were randomized to receive fesoterodine 4 mg PR tablet orally once daily for 12 weeks in active comparator phase. Active comparator phase was followed by safety extension phase, where participants continued to receive fesoterodine 4 mg PR tablet orally once daily for another 12 weeks.
- Cohort 1: Oxybutynin: Participants with body weight >25 kg were randomized to receive oxybutynin ER tablet, at a daily dose in accordance with approved pediatric labeling and accepted practice. Dose titration was done for first 4 weeks. After Week 4, participants remained on the optimized daily dose for next 8 weeks, in active comparator phase.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Fesoterodine 4 mg | Cohort 1: Fesoterodine 4 mg Then 8 mg | Cohort 1: Oxybutynin | Cohort 2: Fesoterodine 2 mg | Cohort 2: Fesoterodine 2 mg Then 4 mg | Total
Number analyzed (Participants) | 42 | 42 | 40 | 28 | 29 | 181
Age, Customized [Count of Participants; unit: Participants]
  >=6-9 Years | 15 | 15 | 15 | 24 | 23 | 92
  >=10-12 Years | 15 | 14 | 13 | 3 | 5 | 50
  >=13-17 Years | 12 | 13 | 12 | 1 | 1 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 22 | 17 | 12 | 19 | 86
  Male | 26 | 20 | 23 | 16 | 10 | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 1 | 0 | 2 | 8
  Not Hispanic or Latino | 39 | 40 | 39 | 28 | 27 | 173
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 14 | 18 | 22 | 16 | 16 | 86
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 0 | 0 | 3
  White | 24 | 24 | 17 | 12 | 11 | 88
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Maximum Cystometric Bladder Capacity at Week 12: Active Comparator Phase/Efficacy Phase
Description: Maximum cystometric bladder capacity (in milliliter) was defined as maximal tolerable cystometric capacity, until voiding or leaking begins or at a pressure of >=40 centimeter (cm) water (H2O).
Time Frame: Baseline, Week 12
Population: Full analysis set included all participants who were randomized in the study and received at least 1 dose of study medication and had provided baseline primary endpoint data.
Measure: Least Squares Mean (95% Confidence Interval); unit: milliliter
Groups:
- Cohort 1, Active Comparator Phase: Fesoterodine 4 mg: Participants with body weight >25 kg were randomized to receive fesoterodine 4 mg PR tablet orally once daily for 12 weeks in active comparator phase.
- Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg: Participants with body weight >25 kg were randomized to receive fesoterodine 4 mg PR tablets orally once daily for first 1 week and if dose was tolerated well, participants received 8 mg PR tablet orally once daily for next 11 weeks in active comparator phase and if dose was not tolerated then participants were withdrawn from the study.
- Cohort 1, Active Comparator Phase: Oxybutynin: Participants with body weight >25 kg were randomized to receive oxybutynin ER tablet, at a daily dose in accordance with approved pediatric labeling and accepted practice. Dose titration was done for first 4 weeks. After Week 4, participants remained on the optimized daily dose for next 8 weeks, in active comparator phase.
- Cohort 2, Efficacy Phase: Fesoterodine 2 mg: Participants with body weight <=25 kg were randomized to receive fesoterodine 2 mg BIC capsule orally once daily for 12 weeks in efficacy phase.
- Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg: Participants with body weight <=25 kg were randomized to receive fesoterodine 2 mg BIC capsule orally once daily for first 1 week and if dose was tolerated well, participants received 4 mg BIC capsule orally once daily for next 11 weeks in efficacy phase and if dose was not tolerated then participants were withdrawn from the study.
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 41 | 41 | 38 | 25 | 28
milliliter | 58.12 [28.84 to 87.39] | 83.36 [54.22 to 112.49] | 87.17 [56.82 to 117.53] | 23.49 [3.03 to 43.95] | 40.17 [20.84 to 59.50]
Statistical Analysis 1: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg; P-value was calculated for change from Baseline at Week 12, based on an analysis of covariance (ANCOVA) model with terms for treatment group, baseline maximum cystometric bladder capacity and baseline weight; Test type: Superiority; p = 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg; P-value was calculated for change from Baseline at Week 12, based on ANCOVA model with terms for treatment group, baseline maximum cystometric bladder capacity and baseline weight; Test type: Superiority; p < .0001, ANCOVA
Statistical Analysis 3: Comparison: Cohort 1, Active Comparator Phase: Oxybutynin; P-value was calculated for change from Baseline at Week 12, based on an ANCOVA model with terms for treatment group, baseline maximum cystometric bladder capacity and baseline weight; Test type: Superiority; p < .0001, ANCOVA
Statistical Analysis 4: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in Least square (LS) Mean = -29.06, 95% CI 2-sided [-71.42 to 13.31]
Statistical Analysis 5: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in LS Mean = -3.82, 95% CI 2-sided [-45.87 to 38.23]

2. Secondary Outcome: Change From Baseline in Detrusor Pressure at Maximum Bladder Capacity at Week 12: Active Comparator Phase/Efficacy Phase
Description: Detrusor pressure (in cm H2O) at maximum urinary bladder capacity was measured using urodynamic testing.
Time Frame: Baseline, Week 12
Population: Full analysis set included all participants who were randomized in the study and received at least 1 dose of study medication and had provided baseline primary endpoint data. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: cm H2O
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 40 | 41 | 38 | 25 | 28
cm H2O | -2.86 [-7.60 to 1.87] | -1.57 [-6.25 to 3.12] | -2.39 [-7.27 to 2.48] | -2.74 [-10.62 to 5.15] | -9.73 [-17.18 to -2.28]
Statistical Analysis 1: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg; P-value was calculated for change from Baseline at Week 12, based on an ANCOVA model with terms for treatment group, baseline detrusor pressure at maximum bladder capacity and baseline weight; Test type: Superiority; p = 0.2334, ANCOVA
Statistical Analysis 2: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.5087, ANCOVA
Statistical Analysis 3: Comparison: Cohort 1, Active Comparator Phase: Oxybutynin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.3333, ANCOVA
Statistical Analysis 4: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in LS Mean = -0.47, 95% CI 2-sided [-7.28 to 6.33]
Statistical Analysis 5: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in LS Mean = 0.82, 95% CI 2-sided [-5.96 to 7.60]

3. Secondary Outcome: Number of Participants With Shift From Baseline at Week 12 in Involuntary Detrusor Contractions (IDC): Active Comparator Phase/Efficacy Phase
Description: In this outcome measure, shift data have been reported using 4 categories: (1) number of participants who did not have IDC at Baseline and at Week 12, (2) number of participants who did not have IDC at Baseline but had IDC at Week 12, (3) number of participants who had IDC at Baseline but no IDC at Week 12, and (4) number of participants who had IDC at Baseline and at Week 12.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 41 | 41 | 38 | 25 | 28
Participants
  Baseline IDC = No; Week 12 IDC = No | 12 | 4 | 6 | 0 | 1
  Baseline IDC = No; Week 12 IDC = Yes | 2 | 1 | 0 | 0 | 0
  Baseline IDC = Yes; Week 12 IDC = No | 9 | 18 | 14 | 6 | 11
  Baseline IDC = Yes; Week 12 IDC = Yes | 18 | 18 | 18 | 19 | 16

4. Secondary Outcome: Change From Baseline in Bladder Volume at First Involuntary Detrusor Contraction (IDC) at Week 12: Active Comparator Phase/Efficacy Phase
Description: Bladder volume (in milliliter) at first IDC was measured using urodynamic testing.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: milliliter
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 26 | 36 | 32 | 25 | 27
milliliter | 30.53 [2.42 to 58.64] | 26.06 [2.19 to 49.92] | 41.31 [15.92 to 66.70] | 23.80 [-1.60 to 49.19] | 31.26 [6.85 to 55.68]
Statistical Analysis 1: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg; P-value was calculated for change from Baseline at Week 12, based on an ANCOVA model with terms for treatment group, baseline bladder volume at first IDC and baseline weight; Test type: Superiority; p = 0.0336, ANCOVA
Statistical Analysis 2: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0327, ANCOVA
Statistical Analysis 3: Comparison: Cohort 1, Active Comparator Phase: Oxybutynin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0017, ANCOVA
Statistical Analysis 4: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in LS Mean = -10.78, 95% CI 2-sided [-48.75 to 27.19]
Statistical Analysis 5: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in LS Mean = -15.25, 95% CI 2-sided [-50.15 to 19.64]

5. Secondary Outcome: Change From Baseline in Bladder Compliance at Week 12: Active Comparator Phase/Efficacy Phase
Description: Bladder compliance was defined as change in bladder volume in milliliter (mL) divided by change in bladder pressure in cm H2O (during the same time when change in bladder volume was estimated).
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mL per cm H2O
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 40 | 40 | 38 | 25 | 28
mL per cm H2O | 6.40 [-0.48 to 13.28] | 5.41 [-1.49 to 12.32] | 11.36 [4.30 to 18.42] | 12.44 [-0.64 to 25.53] | 16.44 [4.08 to 28.80]
Statistical Analysis 1: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg; P-value was calculated for change from Baseline at Week 12, based on an ANCOVA model with terms for treatment group, baseline bladder compliance and baseline weight; Test type: Superiority; p = 0.0679, ANCOVA
Statistical Analysis 2: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.1233, ANCOVA
Statistical Analysis 3: Comparison: Cohort 1, Active Comparator Phase: Oxybutynin; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0019, ANCOVA
Statistical Analysis 4: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in LS Mean = -4.96, 95% CI 2-sided [-14.81 to 4.89]
Statistical Analysis 5: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in LS Mean = -5.95, 95% CI 2-sided [-15.85 to 3.95]

6. Secondary Outcome: Change From Baseline in Mean Number of Micturitions Per 24 Hours at Week 12: Active Comparator Phase/Efficacy Phase
Description: The mean number of micturitions per 24 hours were calculated as the total number of micturitions divided by the total number of diary days collected at the assessment time point. Number of diary days collected at the assessment time point = number of calendar days when the diary was completed on, even if it was not a full 24 hour period. This outcome measure was only calculated for participants with >0 micturitions at Baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: micturitions per 24 hours
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 18 | 21 | 26 | 14 | 17
micturitions per 24 hours | -1.07 [-1.88 to -0.25] | -0.68 [-1.44 to 0.08] | -0.97 [-1.65 to -0.29] | -0.37 [-1.10 to 0.36] | -0.70 [-1.36 to -0.04]
Statistical Analysis 1: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg; P-value was calculated for change from Baseline at Week 12, based on an ANCOVA model with terms for treatment group, baseline number of micturitions per 24 hours and baseline weight; Test type: Superiority; p = 0.0116, ANCOVA
Statistical Analysis 2: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0765, ANCOVA
Statistical Analysis 3: Comparison: Cohort 1, Active Comparator Phase: Oxybutynin; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0061, ANCOVA
Statistical Analysis 4: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in LS Mean = -0.10, 95% CI 2-sided [-1.16 to 0.97]
Statistical Analysis 5: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in LS Mean = 0.28, 95% CI 2-sided [-0.74 to 1.31]

7. Secondary Outcome: Change From Baseline in Mean Number of Catheterizations Per 24 Hours at Week 12: Active Comparator Phase/Efficacy Phase
Description: The mean number of catheterizations per 24 hours were calculated as the total number of catheterizations divided by the total number of diary days collected at the assessment time point. Number of diary days collected at the assessment time point = number of calendar days when the diary was completed on; even if it was not a full 24 hours period. This outcome measure was only calculated for participants with >0 catheterizations at Baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: catheterizations per 24 hours
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 37 | 33 | 31 | 22 | 24
catheterizations per 24 hours | -0.30 [-0.63 to 0.04] | -0.32 [-0.68 to 0.03] | -0.34 [-0.71 to 0.02] | -0.10 [-0.50 to 0.29] | -0.22 [-0.60 to 0.16]
Statistical Analysis 1: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg; P-value was calculated for change from Baseline at Week 12, based on an ANCOVA model with terms for treatment group, baseline number of catheterizations per 24 hours and baseline weight; Test type: Superiority; p = 0.0787, ANCOVA
Statistical Analysis 2: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.0727, ANCOVA
Statistical Analysis 3: Comparison: Cohort 1, Active Comparator Phase: Oxybutynin; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.0666, ANCOVA
Statistical Analysis 4: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in LS Mean = 0.04, 95% CI 2-sided [-0.45 to 0.54]
Statistical Analysis 5: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in LS Mean = 0.02, 95% CI 2-sided [-0.49 to 0.52]

8. Secondary Outcome: Change From Baseline in Mean Number of Micturitions or Catheterizations Per 24 Hours at Week 12: Active Comparator Phase/Efficacy Phase
Description: The mean number of micturitions or catheterizations combined per 24 hours were calculated as the total number of micturitions and catheterizations combined divided by the total number of diary days collected at the assessment point. Number of diary days collected at the assessment time point = number of calendar days when the diary was completed; even if it was not a full 24 hour (hrs) period. This outcome was evaluated in those participants who had micturitions or catheterizations >0 at Baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: micturitions and catheterizations/24 hrs
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 41 | 37 | 38 | 23 | 26
micturitions and catheterizations/24 hrs | -0.61 [-1.08 to -0.14] | -0.60 [-1.09 to -0.11] | -0.75 [-1.24 to -0.26] | -0.24 [-0.67 to 0.19] | -0.28 [-0.68 to 0.12]
Statistical Analysis 1: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg; P-value was calculated for change from Baseline at Week 12, based on an ANCOVA model with terms for treatment group, baseline number of micturitions and catheterizations combined per 24 hours and baseline weight; Test type: Superiority; p = 0.0111, ANCOVA
Statistical Analysis 2: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0171, ANCOVA
Statistical Analysis 3: Comparison: Cohort 1, Active Comparator Phase: Oxybutynin; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0028, ANCOVA
Statistical Analysis 4: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in LS Mean = 0.14, 95% CI 2-sided [-0.53 to 0.82]
Statistical Analysis 5: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in LS Mean = 0.15, 95% CI 2-sided [-0.54 to 0.84]

9. Secondary Outcome: Change From Baseline in Mean Number of Incontinence Episodes Per 24 Hours at Week 12: Active Comparator Phase/Efficacy Phase
Description: The mean number of incontinence episodes per 24 hours were calculated as the total number of incontinence episodes divided by the total number of diary days collected at the assessment time point. Number of diary days collected at the assessment time point = number of calendar days when the diary was completed; even if it was not a full 24 hours period. This outcome measure was only calculated for participants with >0 incontinence episodes at Baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: incontinence episodes per 24 hours
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 33 | 33 | 35 | 22 | 20
incontinence episodes per 24 hours | -0.46 [-0.92 to -0.00] | -0.89 [-1.35 to -0.43] | -1.01 [-1.46 to -0.56] | -0.38 [-0.95 to 0.20] | -0.69 [-1.29 to -0.08]
Statistical Analysis 1: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg; P-value was calculated for change from Baseline at Week 12, based on an ANCOVA model with terms for treatment group, baseline number of incontinence episodes per 24 hours and baseline weight; Test type: Superiority; p = 0.0496, ANCOVA
Statistical Analysis 2: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.0002, ANCOVA
Statistical Analysis 3: Comparison: Cohort 1, Active Comparator Phase: Oxybutynin; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p < .0001, ANCOVA
Statistical Analysis 4: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in LS Mean = 0.55, 95% CI 2-sided [-0.09 to 1.19]
Statistical Analysis 5: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in LS Mean = 0.12, 95% CI 2-sided [-0.52 to 0.77]

10. Secondary Outcome: Change From Baseline in Mean Number of Urgency Episodes Per 24 Hours at Week 12: Active Comparator Phase/Efficacy Phase
Description: The mean number of urgency episodes per 24 hours were calculated as the total number of urgency episodes divided by the total number of diary days collected at the assessment time point. Number of diary days collected at the assessment time point = number of calendar days when the diary was completed; even if it was not a full 24 hours period. Urgency episodes were defined as urgency marked as 'yes' in the diary. This outcome measure was only calculated for participants with >0 urgency episodes at Baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: urgency episodes per 24 hours
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 26 | 18 | 26 | 13 | 9
urgency episodes per 24 hours | -0.62 [-1.18 to -0.06] | -0.50 [-1.17 to 0.17] | -0.14 [-0.70 to 0.42] | -0.23 [-0.84 to 0.38] | -0.62 [-1.35 to 0.12]
Statistical Analysis 1: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg; P-value was calculated for change from Baseline at Week 12, based on an ANCOVA model with terms for treatment group, baseline number of urgency episodes per 24 hours and baseline weight; Test type: Superiority; p = 0.0298, ANCOVA
Statistical Analysis 2: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.1417, ANCOVA
Statistical Analysis 3: Comparison: Cohort 1, Active Comparator Phase: Oxybutynin; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.6219, ANCOVA
Statistical Analysis 4: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in LS Mean = -0.48, 95% CI 2-sided [-1.28 to 0.32]
Statistical Analysis 5: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in LS Mean = -0.36, 95% CI 2-sided [-1.24 to 0.52]

11. Secondary Outcome: Change From Baseline in Mean Volume Voided Per Micturition at Week 12: Active Comparator Phase/Efficacy Phase
Description: The mean voided volume per micturition was calculated as sum of voided volume divided by the total number of micturition episodes with a recorded voided volume greater than 0.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: milliliter per micturition
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 15 | 15 | 20 | 8 | 10
milliliter per micturition | 4.10 [-28.05 to 36.24] | 19.21 [-12.67 to 51.10] | 4.15 [-22.69 to 30.98] | -12.72 [-34.96 to 9.52] | -8.41 [-28.27 to 11.44]
Statistical Analysis 1: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg; P-value was calculated for change from Baseline at Week 12, based on an ANCOVA model with terms for treatment group, baseline mean volume voided per micturition and baseline weight; Test type: Superiority; p = 0.7986, ANCOVA
Statistical Analysis 2: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.2313, ANCOVA
Statistical Analysis 3: Comparison: Cohort 1, Active Comparator Phase: Oxybutynin; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.7571, ANCOVA
Statistical Analysis 4: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in LS Mean = -0.05, 95% CI 2-sided [-42.11 to 42.00]
Statistical Analysis 5: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in LS Mean = 15.07, 95% CI 2-sided [-26.50 to 56.63]

12. Secondary Outcome: Change From Baseline in Mean Volume Voided Per Catheterization at Week 12: Active Comparator Phase/Efficacy Phase
Description: The mean volume per catheterization was calculated as sum of voided volume divided by the total number of catheterization, with a recorded voided volume greater than 0.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: milliliter per catheterization
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 36 | 32 | 28 | 23 | 25
milliliter per catheterization | 29.47 [-1.38 to 60.32] | 47.18 [14.74 to 79.62] | 45.90 [11.24 to 80.55] | 11.50 [-9.87 to 32.88] | 1.74 [-18.76 to 22.23]
Statistical Analysis 1: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg; P-value was calculated for change from Baseline at Week 12, based on an ANCOVA model with terms for treatment group, baseline mean volume voided per catheterization and baseline weight; Test type: Superiority; p = 0.0610, ANCOVA
Statistical Analysis 2: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.0048, ANCOVA
Statistical Analysis 3: Comparison: Cohort 1, Active Comparator Phase: Oxybutynin; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.0100, ANCOVA
Statistical Analysis 4: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in LS Mean = -16.43, 95% CI 2-sided [-63.14 to 30.29]
Statistical Analysis 5: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in LS Mean = 1.28, 95% CI 2-sided [-46.00 to 48.57]

13. Secondary Outcome: Change From Baseline in Mean Volume Voided Per Micturition or Catheterization at Week 12: Active Comparator Phase/Efficacy Phase
Description: The mean voided volume per micturition or catheterization was calculated as sum of voided volume divided by the total number of micturition or catheterization episodes with a recorded voided volume greater than 0. This outcome was evaluated in those participants who had micturitions or catheterizations >0 at Baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mL per micturition or catheterization
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 39 | 38 | 38 | 24 | 28
mL per micturition or catheterization | 18.45 [-11.49 to 48.40] | 55.55 [25.80 to 85.31] | 36.69 [6.95 to 66.43] | 7.12 [-11.87 to 26.11] | -2.65 [-20.22 to 14.92]
Statistical Analysis 1: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg; P-value was calculated for change from Baseline at Week 12, based on an ANCOVA model with terms for treatment group, baseline mean volume voided per micturition or catheterization and baseline weight; Test type: Superiority; p = 0.2246, ANCOVA
Statistical Analysis 2: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0003, ANCOVA
Statistical Analysis 3: Comparison: Cohort 1, Active Comparator Phase: Oxybutynin; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0161, ANCOVA
Statistical Analysis 4: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in LS Mean = -18.24, 95% CI 2-sided [-61.00 to 24.53]
Statistical Analysis 5: Comparison: Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg vs Cohort 1, Active Comparator Phase: Oxybutynin; Test type: Other; Difference in LS Mean = 18.86, 95% CI 2-sided [-22.93 to 60.65]

14. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs): Active Comparator Phase/Efficacy Phase
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important events. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AEs included both all serious and non-serious adverse events.
Time Frame: Baseline up to Week 12
Population: Safety analysis set population for active comparator phase and efficacy phase included all participants of respective cohorts who received at least 1 dose of study medication in the relevant phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 42 | 42 | 40 | 28 | 29
Participants
  Treatment Emergent AEs | 26 | 20 | 30 | 19 | 18
  Treatment Emergent SAEs | 3 | 2 | 1 | 2 | 2

15. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs): Safety Extension Phase
Description: as for outcome 14
Time Frame: Week 12 up to Week 26 (including 2 weeks of follow up after last dose)
Population: Safety analysis set population for safety extension phase included all participants of respective cohorts who received at least 1 dose of study medication in the relevant phase of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1, Safety Extension Phase: Fesoterodine 4 mg: Participants with body weight >25 kg received fesoterodine 4 mg PR tablet orally once daily for 12 weeks in safety extension phase.
- Cohort 1, Safety Extension Phase (SEP): Fesoterodine 8 mg: Participants with body weight >25 kg received fesoterodine 8 mg PR tablet orally once daily for 12 weeks in safety extension phase.
- Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg: Participants with body weight >25 kg who were randomized to receive oxybutynin ER tablet, at a daily dose in accordance with approved pediatric labeling and accepted practice, in active comparator phase; were allocated by investigator to receive fesoterodine 4 mg PR tablet orally once daily for 12 weeks in the safety extension phase.
- Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg Then 8 mg: Participants with body weight >25 kg who were randomized to receive oxybutynin ER tablet, at a daily dose in accordance with approved pediatric labeling and accepted practice, in active comparator phase; were allocated by investigator to receive fesoterodine 4 mg PR tablet orally once daily for first 1 week followed by fesoterodine 8 mg PR tablet orally once daily for another 11 weeks (if the fesoterodine 4 mg dose was well tolerated) in the safety extension phase and if dose was not tolerated participants were withdrawn from the study.
- Cohort 2, Safety Extension Phase: Fesoterodine 2 mg: Participants with body weight <=25 kg received fesoterodine 2 mg BIC capsules orally once daily for 12 weeks in safety extension phase.
- Cohort 2, Safety Extension Phase: Fesoterodine 4 mg: Participants with body weight <=25 kg received fesoterodine 4 mg BIC capsules orally once daily for 12 weeks in safety extension phase.
Arm/Group | Cohort 1, Safety Extension Phase: Fesoterodine 4 mg | Cohort 1, Safety Extension Phase (SEP): Fesoterodine 8 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg Then 8 mg | Cohort 2, Safety Extension Phase: Fesoterodine 2 mg | Cohort 2, Safety Extension Phase: Fesoterodine 4 mg
Number analyzed (Participants) | 30 | 37 | 16 | 20 | 20 | 28
Participants
  Treatment emergent AEs | 14 | 13 | 9 | 11 | 11 | 16
  Treatment emergent SAEs | 0 | 2 | 0 | 0 | 0 | 2

16. Secondary Outcome: Change From Baseline in Visual Acuity at Week 12: Active Comparator Phase/Efficacy Phase
Description: Visual acuity (VA) was assessed using the Snellen method, where logarithm of minimum angle of resolution (logMAR) units were derived from the Snellen ratios. Participants had to read letters from the chart at a distance of 20 feet/6 meter or 4 meter. VA/Snellen ratio = distance between the chart and participant, divided by the distance at which participant was able to see or read chart without impairment; expressed as decimal. logMAR = log10 (1/decimal VA). In this outcome measure data have been reported for right and left eye separately.
Time Frame: Baseline, Week 12
Population: Safety analysis set population for active comparator phase and efficacy phase included all participants of respective cohorts who received at least 1 dose of study medication in the relevant phase. Here, 'Number Analyzed' = participants evaluable for this outcome measure for specified rows.
Measure: Mean (Standard Deviation); unit: logMAR unit
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 42 | 42 | 40 | 28 | 29
logMAR unit
  Right Eye: Baseline: number analyzed (Participants) | 42 | 41 | 40 | 28 | 29
  Right Eye: Baseline | 0.09 (0.16) | 0.11 (0.19) | 0.03 (0.11) | 0.15 (0.21) | 0.10 (0.18)
  Right Eye: Change at Week 12: number analyzed (Participants) | 37 | 40 | 40 | 24 | 29
  Right Eye: Change at Week 12 | 0.01 (0.11) | -0.01 (0.10) | 0.02 (0.18) | 0.03 (0.12) | -0.00 (0.09)
  Left Eye: Baseline | 0.08 (0.16) | 0.10 (0.17) | 0.02 (0.13) | 0.16 (0.21) | 0.14 (0.30)
  Left Eye: Change at Week 12: number analyzed (Participants) | 37 | 41 | 40 | 24 | 29
  Left Eye: Change at Week 12 | 0.00 (0.13) | -0.01 (0.10) | 0.00 (0.13) | -0.02 (0.08) | 0.00 (0.08)

17. Secondary Outcome: Change From Baseline in Visual Acuity at Week 24: Safety Extension Phase
Description: VA was assessed using the Snellen method, where logMAR units were derived from the Snellen ratios. Participants had to read letters from the chart at a distance of 20 feet/6 meter or 4 meter. VA/Snellen ratio = distance between the chart and participant, divided by the distance at which participant was able to see or read chart without impairment; expressed as decimal. logMAR = log10 (1/decimal VA). In this outcome measure data have been reported for right and left eye separately.
Time Frame: Baseline, Week 24
Population: Safety analysis set population for safety extension phase included all participants of respective cohorts who received at least 1 dose of study medication in the relevant phase. Here, 'Number Analyzed' = participants evaluable for this outcome measure for specified rows.
Measure: Mean (Standard Deviation); unit: logMAR unit
Groups:
- Cohort 1, Safety Extension Phase: Fesoterodine 8 mg: Participants with body weight >25 kg received fesoterodine 8 mg PR tablet orally once daily for 12 weeks in safety extension phase.
Arm/Group | Cohort 1, Safety Extension Phase: Fesoterodine 4 mg | Cohort 1, Safety Extension Phase: Fesoterodine 8 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg Then 8 mg | Cohort 2, Safety Extension Phase: Fesoterodine 2 mg | Cohort 2, Safety Extension Phase: Fesoterodine 4 mg
Number analyzed (Participants) | 30 | 37 | 16 | 20 | 20 | 28
logMAR unit
  Right Eye: Change at Week 24: number analyzed (Participants) | 30 | 36 | 16 | 20 | 19 | 28
  Right Eye: Change at Week 24 | 0.04 (0.17) | -0.02 (0.11) | -0.01 (0.05) | 0.02 (0.13) | 0.00 (0.07) | 0.01 (0.11)
  Left Eye: Change at Week 24: number analyzed (Participants) | 30 | 37 | 16 | 20 | 19 | 28
  Left Eye: Change at Week 24 | 0.01 (0.19) | -0.01 (0.11) | 0.00 (0.08) | -0.04 (0.09) | -0.02 (0.07) | 0.03 (0.13)

18. Secondary Outcome: Change From Baseline in Visual Accommodation at Week 12: Active Comparator Phase/Efficacy Phase
Description: The visual accommodation was the distance for each eye at which vision became blurred and was calculated as the mean of triplicate measurements. The participants focused on a single letter of the 20/40 line of an eye chart and chart was moved slowly towards the participant until letter was blurred. At this point, the distance from eye to letter was measured for each eye. In this outcome measure data have been reported for right and left eye separately.
Time Frame: Baseline, Week 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 42 | 42 | 40 | 28 | 29
centimeter
  Right Eye: Baseline: number analyzed (Participants) | 38 | 39 | 39 | 26 | 28
  Right Eye: Baseline | 11.88 (7.39) | 15.94 (18.64) | 9.59 (5.05) | 9.67 (16.71) | 8.17 (6.89)
  Right Eye: Change at Week 12: number analyzed (Participants) | 33 | 38 | 39 | 22 | 28
  Right Eye: Change at Week 12 | 1.74 (7.45) | 7.77 (45.53) | 0.50 (4.64) | -1.04 (6.79) | 1.02 (3.89)
  Left Eye: Baseline: number analyzed (Participants) | 39 | 40 | 39 | 26 | 27
  Left Eye: Baseline | 12.31 (8.67) | 15.83 (17.85) | 9.69 (5.13) | 8.81 (14.89) | 8.04 (7.17)
  Left Eye: Change at Week 12: number analyzed (Participants) | 34 | 39 | 39 | 22 | 27
  Left Eye: Change at Week 12 | 0.27 (4.29) | 5.79 (36.75) | 0.81 (4.78) | -1.45 (9.60) | 0.90 (3.38)

19. Secondary Outcome: Change From Baseline in Visual Accommodation at Week 24: Safety Extension Phase
Description: The visual accommodation is the distance for each eye at which vision became blurred and was calculated as the mean of triplicate measurements. The participants focused on a single letter of the 20/40 line of an eye chart and chart was moved slowly towards the participant until letter was blurred. At this point, the distance from eye to letter was measured for each eye. In this outcome measure data have been reported for right and left eye separately.
Time Frame: Baseline, Week 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Cohort 1, Safety Extension Phase: Fesoterodine 4 mg | Cohort 1, Safety Extension Phase: Fesoterodine 8 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg Then 8 mg | Cohort 2, Safety Extension Phase: Fesoterodine 2 mg | Cohort 2, Safety Extension Phase: Fesoterodine 4 mg
Number analyzed (Participants) | 30 | 37 | 16 | 20 | 20 | 28
centimeter
  Right Eye: Change at Week 24: number analyzed (Participants) | 27 | 34 | 16 | 20 | 18 | 27
  Right Eye: Change at Week 24 | 0.73 (5.47) | 4.33 (28.89) | 1.50 (4.80) | 0.50 (4.30) | -1.35 (13.03) | 0.96 (4.38)
  Left Eye: Change at Week 24: number analyzed (Participants) | 28 | 35 | 16 | 20 | 18 | 26
  Left Eye: Change at Week 24 | 0.90 (5.85) | 3.79 (29.81) | 1.66 (6.25) | 0.58 (4.53) | 0.43 (11.53) | 1.12 (4.20)

20. Secondary Outcome: Change From Baseline in Child Behavior Checklist (CBCL) T Score (Derived Score) at Week 12: Active Comparator Phase/Efficacy Phase
Description: CBCL: 120 items questionnaire answered by parent/caregiver of child to assess a child's behavioral, emotional problems. Scale for each item: 0= not true, 1= somewhat/sometimes true, 2= very true/often true. Out of 120 items, 103 were categorized into 8 domains; aggressive behavior, anxious/depressed, attention problems, rule-breaking behavior, social problems, somatic complaints, thought problems, withdrawn. Summary scores: Internalizing problems=anxious/depressed + withdrawn + somatic complaints; Externalizing problems=rule-breaking + aggressive behavior. Total problems=8 domains + other 17 items. Raw scores for each domain, summary and total problems=sum of scores of related items. Using Assessment Data Manager (ADM) tool raw scores transformed/derived into standard T-scores, range: each domain=50 to 100, internalizing problems=34 to 100, externalizing problems=33 to 100, total problems=24 to 100. Lower T-score for each 8 domains, 2 summary and total problems scores=better outcomes.
Time Frame: Baseline, Week 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 42 | 42 | 40 | 28 | 29
T score
  Aggressive behavior: Baseline: number analyzed (Participants) | 42 | 41 | 40 | 28 | 29
  Aggressive behavior: Baseline | 53.86 (5.67) | 54.32 (5.88) | 54.58 (5.75) | 54.9 (5.25) | 52.8 (4.48)
  Aggressive behavior: Change at Week 12: number analyzed (Participants) | 37 | 40 | 39 | 24 | 29
  Aggressive behavior: Change at Week 12 | -1.03 (3.17) | -0.95 (3.71) | -1.28 (2.77) | -1.29 (3.58) | -0.03 (2.96)
  Anxious/depressed: Baseline: number analyzed (Participants) | 42 | 41 | 40 | 28 | 29
  Anxious/depressed: Baseline | 56.07 (6.99) | 57.00 (8.26) | 56.75 (7.32) | 55.5 (6.58) | 56.3 (6.55)
  Anxious/depressed: Change at Week 12: number analyzed (Participants) | 37 | 40 | 39 | 24 | 29
  Anxious/depressed: Change at Week 12 | -1.73 (3.05) | -1.38 (5.25) | -1.92 (4.66) | -0.79 (4.55) | -3.21 (5.27)
  Attention problems: Baseline: number analyzed (Participants) | 42 | 41 | 40 | 28 | 29
  Attention problems: Baseline | 56.29 (5.32) | 56.66 (7.47) | 56.30 (5.68) | 55.4 (5.06) | 55.3 (5.74)
  Attention problems: Change at week 12: number analyzed (Participants) | 37 | 40 | 39 | 24 | 29
  Attention problems: Change at week 12 | -1.97 (3.79) | -1.40 (4.30) | -1.28 (3.69) | -1.29 (3.61) | -1.45 (3.41)
  Rule-breaking behavior: Baseline: number analyzed (Participants) | 42 | 41 | 40 | 28 | 29
  Rule-breaking behavior: Baseline | 53.26 (3.52) | 53.80 (5.53) | 53.43 (4.96) | 54.5 (4.96) | 52.3 (3.74)
  Rule-breaking behavior: Change at Week 12: number analyzed (Participants) | 37 | 40 | 39 | 24 | 29
  Rule-breaking behavior: Change at Week 12 | -0.92 (2.99) | -0.88 (3.91) | -0.72 (2.76) | -1.71 (4.84) | -0.10 (2.19)
  Social problems : Baseline: number analyzed (Participants) | 42 | 41 | 40 | 28 | 29
  Social problems : Baseline | 57.52 (5.42) | 58.54 (9.43) | 57.95 (7.90) | 57.9 (6.66) | 55.8 (5.90)
  Social problems : Change at Week 12: number analyzed (Participants) | 37 | 40 | 39 | 24 | 29
  Social problems : Change at Week 12 | -1.35 (3.90) | -2.55 (4.74) | -0.67 (3.73) | -2.21 (4.38) | -1.10 (3.41)
  Somatic complaints: Baseline: number analyzed (Participants) | 42 | 41 | 40 | 28 | 29
  Somatic complaints: Baseline | 61.14 (6.24) | 60.46 (8.73) | 60.58 (8.44) | 57.1 (6.47) | 58.4 (6.55)
  Somatic complaints: Change at Week 12: number analyzed (Participants) | 37 | 40 | 39 | 24 | 29
  Somatic complaints: Change at Week 12 | -0.46 (5.99) | -1.28 (6.35) | -0.87 (7.16) | -0.38 (3.97) | -1.69 (5.90)
  Thought problems: Baseline: number analyzed (Participants) | 42 | 41 | 40 | 28 | 29
  Thought problems: Baseline | 55.00 (6.19) | 53.54 (5.93) | 56.73 (7.64) | 51.9 (2.81) | 54.9 (5.60)
  Thought problems: Change at Week 12: number analyzed (Participants) | 37 | 40 | 39 | 24 | 29
  Thought problems: Change at Week 12 | -0.92 (4.69) | -0.48 (4.25) | -1.59 (3.65) | -0.42 (1.67) | -1.38 (5.42)
  Withdrawn: Baseline: number analyzed (Participants) | 42 | 41 | 40 | 28 | 29
  Withdrawn: Baseline | 54.60 (5.17) | 57.54 (8.34) | 58.25 (7.93) | 55.7 (5.96) | 55.0 (7.11)
  Withdrawn: Change at Week 12: number analyzed (Participants) | 37 | 40 | 39 | 24 | 29
  Withdrawn: Change at Week 12 | 0.35 (4.70) | -1.25 (5.13) | -1.92 (5.08) | -1.75 (3.97) | -0.59 (4.48)
  Externalizing: Baseline: number analyzed (Participants) | 42 | 41 | 40 | 28 | 29
  Externalizing: Baseline | 49.48 (8.68) | 49.46 (10.00) | 50.10 (9.73) | 51.1 (9.83) | 48.0 (7.84)
  Externalizing: Change at Week 12: number analyzed (Participants) | 37 | 40 | 39 | 24 | 29
  Externalizing: Change at Week 12 | -2.08 (5.26) | -2.33 (5.28) | -1.95 (4.62) | -2.63 (4.72) | -1.45 (4.56)
  Internalizing: Baseline: number analyzed (Participants) | 42 | 41 | 40 | 28 | 29
  Internalizing: Baseline | 56.45 (8.06) | 55.93 (12.84) | 57.25 (11.00) | 53.9 (10.34) | 54.6 (10.14)
  Internalizing: Change at Week 12: number analyzed (Participants) | 37 | 40 | 39 | 24 | 29
  Internalizing: Change at Week 12 | -2.14 (6.46) | -2.35 (6.98) | -3.05 (7.12) | -1.96 (6.53) | -3.52 (6.38)
  Total Problems: Baseline: number analyzed (Participants) | 42 | 41 | 40 | 28 | 29
  Total Problems: Baseline | 55.05 (8.20) | 53.61 (11.98) | 55.45 (10.28) | 53.4 (10.70) | 52.7 (9.37)
  Total Problems: Change at Week 12 | -2.51 (4.63) | -3.23 (5.45) | -2.36 (4.68) | -2.17 (5.05) | -3.38 (4.55)

21. Secondary Outcome: Change From Baseline in Child Behavior Checklist (CBCL) T Score (Derived Score) at Week 24: Safety Extension Phase
Description: as for outcome 20
Time Frame: Baseline, Week 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Cohort 1, Safety Extension Phase: Fesoterodine 4 mg | Cohort 1, Safety Extension Phase: Fesoterodine 8 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg Then 8 mg | Cohort 2, Safety Extension Phase: Fesoterodine 2 mg | Cohort 2, Safety Extension Phase: Fesoterodine 4 mg
Number analyzed (Participants) | 30 | 37 | 16 | 20 | 20 | 28
T score
  Aggressive behavior: Change at Week 24: number analyzed (Participants) | 29 | 36 | 16 | 20 | 20 | 28
  Aggressive behavior: Change at Week 24 | -1.59 (3.85) | -1.31 (4.57) | -1.25 (3.40) | -2.40 (4.89) | -1.70 (3.40) | -1.86 (3.63)
  Anxious/depressed: Change at Week 24: number analyzed (Participants) | 29 | 36 | 16 | 20 | 20 | 28
  Anxious/depressed: Change at Week 24 | -3.45 (4.86) | -2.31 (5.64) | -1.50 (3.76) | -3.25 (5.66) | -2.60 (5.24) | -3.89 (4.95)
  Attention problems: Change at Week 24: number analyzed (Participants) | 29 | 36 | 16 | 20 | 20 | 28
  Attention problems: Change at Week 24 | -2.21 (3.99) | -2.64 (5.72) | -3.38 (4.65) | -1.70 (3.01) | -1.50 (3.15) | -1.71 (3.29)
  Rule-breaking behavior: Change at Week 24: number analyzed (Participants) | 29 | 36 | 16 | 20 | 20 | 28
  Rule-breaking behavior: Change at Week 24 | -1.59 (3.62) | -1.47 (5.12) | -1.31 (4.01) | -0.90 (2.36) | -2.15 (3.17) | -0.36 (2.63)
  Social problems : Change at Week 24: number analyzed (Participants) | 29 | 36 | 16 | 20 | 20 | 28
  Social problems : Change at Week 24 | -2.83 (4.12) | -2.56 (4.15) | -3.19 (5.79) | -2.65 (3.28) | -3.90 (4.35) | -2.36 (4.17)
  Somatic complaints: Change at Week 24: number analyzed (Participants) | 29 | 36 | 16 | 20 | 20 | 28
  Somatic complaints: Change at Week 24 | -4.38 (6.59) | -2.64 (6.58) | -1.69 (9.20) | -1.50 (5.82) | -0.60 (3.12) | -1.96 (6.77)
  Thought problems: Change at Week 24: number analyzed (Participants) | 29 | 36 | 16 | 20 | 20 | 28
  Thought problems: Change at Week 24 | -3.10 (5.45) | -1.03 (4.52) | -3.25 (6.62) | -2.30 (3.50) | -1.40 (3.00) | -1.75 (3.99)
  Withdrawn: Change at Week 24: number analyzed (Participants) | 29 | 36 | 16 | 20 | 20 | 28
  Withdrawn: Change at Week 24 | -0.69 (4.33) | -1.50 (5.98) | -2.19 (3.90) | -4.35 (5.24) | -1.80 (5.43) | -0.43 (3.75)
  Externalizing: Change at Week 24: number analyzed (Participants) | 29 | 36 | 16 | 20 | 20 | 28
  Externalizing: Change at Week 24 | -5.21 (8.20) | -2.89 (7.06) | -1.81 (5.42) | -4.15 (7.44) | -4.20 (5.15) | -4.21 (6.86)
  Internalizing: Change at Week 24: number analyzed (Participants) | 29 | 36 | 16 | 20 | 20 | 28
  Internalizing: Change at Week 24 | -7.69 (7.46) | -4.14 (7.62) | -3.25 (8.10) | -5.35 (7.21) | -4.40 (6.21) | -4.32 (6.70)
  Total Problems: Change at Week 24 | -7.03 (7.77) | -4.44 (6.57) | -3.69 (6.74) | -4.90 (4.78) | -5.20 (4.32) | -5.25 (6.22)

22. Secondary Outcome: Change From Baseline in Child Behavior Checklist Total Score (Raw Score) at Week 12: Active Comparator Phase/Efficacy Phase
Description: CBCL: It consisted of 120 items on behavior and emotional problems. Parent/caregiver of child answered 120 items, each on scale: 0= not true, 1= somewhat/sometimes true, 2= very/often true. 103 items were classified in 8 domains: aggressive behavior: total score range (TSR)= 0 to 36, anxious/depressed: TSR= 0 to 26, attention problems: TSR= 0 to 20, rule-breaking behavior: TSR= 0 to 34, social problems: TSR= 0 to 22, somatic complaints: TSR= 0 to 22, thought problems: TSR= 0 to 30, withdrawn (TSR)= 0 to 16. Rule-breaking and aggressive behavior summarized to externalizing problems with a TSR= 0 to 70. Anxious/depressed, withdrawn, somatic complaints summarized to internalizing problems with a TSR= 0 to 64. All 103 items of 8 domains and other 17 remaining items were combined to give total problems TSR = 0 to 240. TSR for each domain, summary and total problems was sum of scores of related items respectively. Lower scores for each domain, summary and total problems= better outcomes.
Time Frame: Baseline, Week 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 42 | 42 | 40 | 28 | 29
units on a scale
  Aggressive behavior: Baseline: number analyzed (Participants) | 42 | 41 | 40 | 28 | 29
  Aggressive behavior: Baseline | 4.19 (4.39) | 4.66 (4.46) | 4.88 (4.35) | 5.1 (3.95) | 3.5 (3.37)
  Aggressive behavior: Change at Week 12: number analyzed (Participants) | 37 | 40 | 39 | 24 | 29
  Aggressive behavior: Change at Week 12 | -0.62 (2.35) | -0.90 (2.56) | -0.97 (2.08) | -0.92 (2.39) | -0.17 (1.85)
  Anxious/depressed: Baseline: number analyzed (Participants) | 42 | 41 | 40 | 28 | 29
  Anxious/depressed: Baseline | 3.83 (3.33) | 4.20 (4.06) | 4.10 (3.53) | 3.8 (3.15) | 4.0 (3.35)
  Anxious/depressed: Change at Week 12: number analyzed (Participants) | 37 | 40 | 39 | 24 | 29
  Anxious/depressed: Change at Week 12 | -0.97 (1.46) | -0.73 (2.43) | -1.05 (2.26) | -0.58 (2.28) | -1.48 (2.43)
  Attention problems: Baseline: number analyzed (Participants) | 42 | 41 | 40 | 28 | 29
  Attention problems: Baseline | 4.79 (3.18) | 4.49 (4.11) | 4.85 (3.33) | 4.2 (2.78) | 3.9 (3.11)
  Attention problems: Change at Week 12: number analyzed (Participants) | 37 | 40 | 39 | 24 | 29
  Attention problems: Change at Week 12 | -1.05 (2.25) | -0.73 (2.16) | -0.77 (2.03) | -0.71 (1.90) | -0.83 (1.63)
  Rule-breaking behavior: Baseline: number analyzed (Participants) | 42 | 41 | 40 | 28 | 29
  Rule-breaking behavior: Baseline | 1.64 (1.48) | 1.66 (1.98) | 1.70 (1.87) | 1.9 (1.63) | 1.0 (1.30)
  Rule-breaking behavior: Change at Week 12: number analyzed (Participants) | 37 | 40 | 39 | 24 | 29
  Rule-breaking behavior: Change at Week 12 | -0.43 (1.09) | -0.30 (1.36) | -0.38 (0.99) | -0.63 (1.56) | 0.52 (3.45)
  Social problems: Baseline: number analyzed (Participants) | 42 | 41 | 40 | 28 | 29
  Social problems: Baseline | 3.60 (2.30) | 4.07 (4.12) | 3.80 (3.36) | 3.9 (2.99) | 3.2 (2.64)
  Social problems: Change at Week 12: number analyzed (Participants) | 37 | 40 | 39 | 24 | 29
  Social problems: Change at Week 12 | -0.54 (1.54) | -1.13 (2.09) | -0.26 (1.57) | -0.83 (1.86) | -0.62 (1.52)
  Somatic complaints: Baseline: number analyzed (Participants) | 42 | 41 | 40 | 28 | 29
  Somatic complaints: Baseline | 3.40 (2.18) | 3.46 (3.26) | 3.40 (3.23) | 2.1 (1.93) | 2.6 (2.16)
  Somatic complaints: Change at Week 12: number analyzed (Participants) | 37 | 40 | 39 | 24 | 29
  Somatic complaints: Change at Week 12 | -0.05 (2.26) | -0.53 (2.44) | -0.51 (2.64) | -0.04 (1.55) | -0.55 (2.03)
  Thought problems: Baseline: number analyzed (Participants) | 42 | 41 | 40 | 28 | 29
  Thought problems: Baseline | 2.05 (2.23) | 1.46 (2.34) | 2.58 (2.92) | 1.0 (1.04) | 2.0 (1.79)
  Thought problems: Change at Week 12: number analyzed (Participants) | 37 | 40 | 39 | 24 | 29
  Thought problems: Change at Week 12 | -0.46 (1.69) | -0.10 (1.37) | -0.51 (1.30) | -0.21 (0.72) | -0.45 (1.64)
  Withdrawn: Baseline: number analyzed (Participants) | 42 | 41 | 40 | 28 | 29
  Withdrawn: Baseline | 1.52 (1.77) | 2.49 (2.78) | 2.75 (2.66) | 1.7 (1.81) | 1.6 (2.26)
  Withdrawn: Change at Week 12: number analyzed (Participants) | 37 | 40 | 39 | 24 | 29
  Withdrawn: Change at Week 12 | 0.14 (1.44) | -0.35 (1.59) | -0.64 (1.77) | -0.50 (1.10) | -0.17 (1.39)
  Externalizing: Baseline: number analyzed (Participants) | 42 | 41 | 40 | 28 | 29
  Externalizing: Baseline | 5.83 (5.23) | 6.32 (6.14) | 6.53 (5.87) | 6.9 (5.16) | 4.5 (4.32)
  Externalizing: Change at Week 12: number analyzed (Participants) | 37 | 40 | 39 | 24 | 29
  Externalizing: Change at Week 12 | -1.05 (2.85) | -1.20 (3.42) | -1.31 (2.30) | -1.54 (3.50) | -0.31 (2.33)
  Internalizing: Baseline: number analyzed (Participants) | 42 | 41 | 40 | 28 | 29
  Internalizing: Baseline | 8.76 (5.56) | 10.15 (8.64) | 10.25 (7.02) | 7.5 (5.61) | 8.2 (6.13)
  Internalizing: Change at Week 12: number analyzed (Participants) | 37 | 40 | 39 | 24 | 29
  Internalizing: Change at Week 12 | -0.89 (3.62) | -1.70 (5.16) | -2.21 (4.35) | -1.13 (3.85) | -2.21 (3.91)
  Total Problems: Baseline: number analyzed (Participants) | 42 | 41 | 40 | 28 | 29
  Total Problems: Baseline | 31.52 (16.84) | 31.88 (23.78) | 34.18 (22.16) | 29.5 (17.41) | 27.0 (16.59)
  Total Problems: Change at Week 12: number analyzed (Participants) | 37 | 40 | 39 | 24 | 29
  Total Problems: Change at Week 12 | -4.92 (8.73) | -5.83 (12.16) | -5.85 (9.77) | -5.33 (8.29) | -5.10 (7.41)

23. Secondary Outcome: Change From Baseline in Child Behavior Checklist Total Score (Raw Score) at Week 24: Safety Extension Phase
Description: as for outcome 22
Time Frame: Baseline, Week 24
Population: Safety analysis set population for safety extension phase: all participants of respective cohorts who received at least 1 dose of study medication in the relevant phase. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1, Safety Extension Phase: Fesoterodine 4 mg | Cohort 1, Safety Extension Phase: Fesoterodine 8 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg Then 8 mg | Cohort 2, Safety Extension Phase: Fesoterodine 2 mg | Cohort 2, Safety Extension Phase: Fesoterodine 4 mg
Number analyzed (Participants) | 29 | 36 | 16 | 20 | 20 | 28
units on a scale
  Aggressive behavior: Change at Week 24 | -1.34 (2.92) | -1.17 (3.10) | -0.81 (2.43) | -1.75 (3.58) | -1.40 (2.41) | -1.57 (2.70)
  Anxious/depressed: Change at Week 24 | -1.93 (2.22) | -1.28 (2.42) | -1.06 (1.88) | -1.60 (2.48) | -1.70 (2.36) | -1.75 (2.34)
  Attention problems: Change at Week 24 | -1.41 (2.31) | -1.36 (2.77) | -1.94 (2.35) | -1.25 (1.77) | -1.15 (1.76) | -0.89 (1.69)
  Rule-breaking behavior: Change at Week 24 | -0.62 (1.29) | -0.50 (1.65) | -0.50 (1.21) | -0.55 (0.94) | -0.80 (1.01) | -0.18 (0.94)
  Social problems: Change at Week 24 | -1.28 (1.53) | -1.19 (1.97) | -1.13 (2.33) | -1.20 (1.36) | -1.65 (1.81) | -1.14 (1.74)
  Somatic complaints: Change at Week 24 | -1.34 (2.22) | -0.89 (2.38) | -0.88 (3.32) | -0.45 (1.73) | -0.15 (0.88) | -0.68 (2.04)
  Thought problems: Change at Week 24 | -1.31 (1.95) | -0.36 (1.40) | -1.06 (2.14) | -0.90 (1.21) | -0.65 (1.04) | -0.64 (1.28)
  Withdrawn: Change at Week 24 | -0.24 (1.43) | -0.44 (2.01) | -0.69 (1.35) | -1.35 (1.66) | -0.45 (1.50) | -0.14 (1.04)
  Externalizing: Change at Week 24 | -1.97 (3.50) | -1.67 (4.27) | -1.19 (3.23) | -2.30 (4.03) | -2.20 (2.84) | -1.79 (3.28)
  Internalizing: Change at Week 24 | -3.52 (4.00) | -2.61 (4.95) | -2.63 (4.65) | -3.40 (4.68) | -2.30 (3.64) | -2.57 (3.63)
  Total Problems: Change at Week 24 | -10.90 (11.98) | -8.58 (12.86) | -9.00 (13.45) | -10.10 (10.47) | -9.45 (7.93) | -8.39 (10.22)

24. Secondary Outcome: Change From Baseline in Time to Completion Assessment of Grooved Pegboard Test, 10 Pegs Group at Week 12: Active Comparator Phase/Efficacy Phase
Description: The grooved pegboard test was a manipulative dexterity test that assessed psychomotor speed, fine motor control, and rapid-visual motor coordination. It consisted of a small board of 25 holes with randomly positioned slots. Pegs with a key along one side must be rotated to match the hole before they can be inserted. In this outcome measure participants were asked to insert 10 grooved pegs into the holes within the given time limit (up to 300 seconds). The task needs to be completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand. Time taken to complete the test was inversely correlated to the cognitive ability.
Time Frame: Baseline, Week 12
Population: Safety analysis set population for active comparator phase and efficacy phase analyzed. 10-peg assessment was done only in participants below age of 9 years. "Overall Number of Participants Analyzed": participants evaluable for this outcome measure, "Number Analyzed": participants evaluable for specified rows. There was 1 participant who inadvertently did the 10-peg test with non-dominant hand and 25-peg test with dominant hand. This participant was counted in both 10 peg and 25 peg assessment.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 9 | 9 | 7 | 18 | 21
seconds
  Dominant hand: Baseline: number analyzed (Participants) | 9 | 8 | 7 | 18 | 20
  Dominant hand: Baseline | 61.11 (31.66) | 56.50 (32.09) | 46.43 (16.28) | 69.56 (58.52) | 52.20 (31.06)
  Dominant hand: Change at Week 12: number analyzed (Participants) | 7 | 7 | 6 | 15 | 19
  Dominant hand: Change at Week 12 | -7.71 (11.06) | 10.14 (37.18) | -5.33 (6.15) | -11.20 (41.11) | -10.26 (27.21)
  Non-dominant hand: Baseline: number analyzed (Participants) | 9 | 9 | 7 | 17 | 21
  Non-dominant hand: Baseline | 80.44 (41.45) | 114.00 (89.43) | 48.00 (15.14) | 91.29 (110.76) | 76.29 (76.71)
  Non-dominant hand: Change at Week 12: number analyzed (Participants) | 7 | 6 | 6 | 14 | 20
  Non-dominant hand: Change at Week 12 | -21.71 (25.44) | 15.33 (49.28) | -2.00 (12.25) | -19.36 (81.03) | -3.25 (22.53)

25. Secondary Outcome: Change From Baseline in Time to Completion Assessment of Grooved Pegboard Test, 10 Pegs Group at Week 24: Safety Extension Phase
Description: as for outcome 24
Time Frame: Baseline, Week 24
Population: Safety analysis set population for active comparator phase and efficacy phase analyzed. 10-peg assessment was done only in participants below age of 9 years. Here, "Overall Number of Participants Analyzed": participants evaluable for this outcome measure and "Number Analyzed": participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cohort 1, Safety Extension Phase: Fesoterodine 4 mg | Cohort 1, Safety Extension Phase: Fesoterodine 8 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg Then 8 mg | Cohort 2, Safety Extension Phase: Fesoterodine 2 mg | Cohort 2, Safety Extension Phase: Fesoterodine 4 mg
Number analyzed (Participants) | 3 | 7 | 2 | 3 | 15 | 19
seconds
  Dominant hand: Change at Week 24: number analyzed (Participants) | 3 | 7 | 2 | 3 | 15 | 18
  Dominant hand: Change at Week 24 | -11.33 (9.07) | -3.71 (22.94) | -2.00 (8.49) | -6.33 (3.06) | -7.07 (6.80) | -15.00 (28.54)
  Non-dominant hand: Change at Week 24: number analyzed (Participants) | 3 | 6 | 2 | 3 | 14 | 19
  Non-dominant hand: Change at Week 24 | -2.00 (13.75) | -4.00 (29.09) | 1.50 (10.61) | -11.00 (5.00) | -9.14 (14.33) | -18.47 (38.13)

26. Secondary Outcome: Change From Baseline in Time to Completion Assessment of Grooved Pegboard Test, 25 Pegs Group at Week 12: Active Comparator Phase/Efficacy Phase
Description: The grooved pegboard test was a manipulative dexterity test that assessed psychomotor speed, fine motor control, and rapid-visual motor coordination. It consisted of a small board of 25 holes with randomly positioned slots. Pegs with a key along one side must be rotated to match the hole before they can be inserted. In this outcome measure participants were asked to insert 25 grooved pegs into the holes within the given time limit (up to 300 seconds). The task needs to be completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand. Time taken to complete the test was inversely correlated to the cognitive ability.
Time Frame: Baseline, Week 12
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 33 | 34 | 33 | 10 | 9
seconds
  Dominant hand: Baseline | 88.85 (24.22) | 92.15 (40.51) | 82.64 (24.32) | 106.7 (64.07) | 124.7 (71.99)
  Dominant hand: Change at Week 12: number analyzed (Participants) | 30 | 33 | 33 | 8 | 9
  Dominant hand: Change at Week 12 | -5.40 (10.43) | -8.88 (20.76) | 1.21 (11.87) | -14.38 (25.90) | -18.44 (32.23)
  Non-dominant hand: Baseline: number analyzed (Participants) | 33 | 32 | 33 | 10 | 8
  Non-dominant hand: Baseline | 110.61 (59.63) | 109.00 (49.75) | 92.94 (25.05) | 130.30 (83.58) | 126.1 (48.93)
  Non-dominant hand: Change at Week 12: number analyzed (Participants) | 30 | 31 | 33 | 8 | 8
  Non-dominant hand: Change at Week 12 | -9.10 (19.94) | -4.10 (10.79) | -1.97 (14.00) | -13.50 (18.81) | -12.50 (20.30)

27. Secondary Outcome: Change From Baseline in Time to Completion Assessment of Grooved Pegboard Test, 25 Pegs Group at Week 24: Safety Extension Phase
Description: as for outcome 26
Time Frame: Baseline, Week 24
Population: Safety analysis set population for active comparator phase and efficacy phase analyzed. 25-peg assessment was done only in participants of age 9 years and above. Here, "Overall Number of Participants Analyzed": participants evaluable for this outcome measure and "Number Analyzed": participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cohort 1, Safety Extension Phase: Fesoterodine 4 mg | Cohort 1, Safety Extension Phase: Fesoterodine 8 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg Then 8 mg | Cohort 2, Safety Extension Phase: Fesoterodine 2 mg | Cohort 2, Safety Extension Phase: Fesoterodine 4 mg
Number analyzed (Participants) | 25 | 30 | 14 | 16 | 5 | 9
seconds
  Dominant hand: Change at Week 24 | -8.20 (11.67) | -12.27 (18.28) | -5.71 (9.55) | -7.00 (13.25) | -38.20 (31.67) | -17.00 (33.16)
  Non-dominant hand: Change at Week 24: number analyzed (Participants) | 25 | 28 | 14 | 15 | 5 | 8
  Non-dominant hand: Change at Week 24 | -9.24 (15.79) | -8.46 (10.42) | -3.79 (11.89) | -11.87 (14.15) | -38.00 (29.35) | -15.50 (29.11)

28. Secondary Outcome: Change From Baseline in Number of Pegs Dropped Assessment of Grooved Pegboard Test, 10 Pegs Group at Week 12: Active Comparator Phase/Efficacy Phase
Description: The grooved pegboard test was a manipulative dexterity test that assessed psychomotor speed, fine motor control, and rapid-visual motor coordination. It consisted of a small board of 25 holes with randomly positioned slots. Pegs with a key along one side must be rotated to match the hole before they can be inserted. Participants were asked to insert 10 grooved pegs into the holes within the given time limit (up to 300 seconds). In this outcome measure number of pegs dropped while putting in the holes were measured. The task needs to be completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand.
Time Frame: Baseline, Week 12
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: pegs
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 9 | 9 | 7 | 18 | 21
pegs
  Dominant hand: Baseline: number analyzed (Participants) | 9 | 8 | 7 | 18 | 20
  Dominant hand: Baseline | 0.11 (0.33) | 0.75 (1.75) | 0.29 (0.49) | 0.39 (1.24) | 0.10 (0.45)
  Dominant hand: Change at Week 12: number analyzed (Participants) | 7 | 7 | 6 | 15 | 19
  Dominant hand: Change at Week 12 | 0.29 (0.76) | 0.57 (1.13) | -0.17 (0.75) | 0.00 (1.77) | 0.05 (0.52)
  Non-dominant hand: Baseline: number analyzed (Participants) | 9 | 9 | 7 | 17 | 21
  Non-dominant hand: Baseline | 0.44 (0.53) | 1.22 (2.28) | 0.00 (0.00) | 0.35 (0.86) | 0.76 (2.26)
  Non-dominant hand: Change at Week 12: number analyzed (Participants) | 7 | 6 | 6 | 14 | 20
  Non-dominant hand: Change at Week 12 | 0.43 (1.27) | 1.00 (2.00) | 0.17 (0.41) | 0.00 (0.68) | 0.60 (3.45)

29. Secondary Outcome: Change From Baseline in Number of Pegs Dropped Assessment of Grooved Pegboard Test, 10 Pegs Group at Week 24: Safety Extension Phase
Description: as for outcome 28
Time Frame: Baseline, Week 24
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: pegs
Groups:
- Cohort 1,SEP: Oxybutynin Then Fesoterodine 8 mg: Participants with body weight >25 kg who were randomized to receive oxybutynin 5 mg ER tablets orally once daily in active comparator phase, were allocated by investigator to receive fesoterodine 8 mg for 12 weeks in safety extension phase.
Arm/Group | Cohort 1, Safety Extension Phase: Fesoterodine 4 mg | Cohort 1, Safety Extension Phase: Fesoterodine 8 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg | Cohort 1,SEP: Oxybutynin Then Fesoterodine 8 mg | Cohort 2, Safety Extension Phase: Fesoterodine 2 mg | Cohort 2, Safety Extension Phase: Fesoterodine 4 mg
Number analyzed (Participants) | 3 | 7 | 2 | 3 | 15 | 19
pegs
  Dominant hand: Change at week 24: number analyzed (Participants) | 3 | 7 | 2 | 3 | 15 | 18
  Dominant hand: Change at week 24 | 0.33 (0.58) | 0.43 (0.79) | 0.00 (0.00) | -0.33 (0.58) | -0.27 (1.39) | -0.06 (0.54)
  Non-dominant hand: Change at week 24: number analyzed (Participants) | 3 | 6 | 2 | 3 | 14 | 19
  Non-dominant hand: Change at week 24 | 1.33 (2.31) | 0.00 (1.10) | 0.50 (0.71) | 0.00 (0.00) | -0.36 (0.74) | 0.11 (3.45)

30. Secondary Outcome: Change From Baseline in Number of Pegs Dropped Assessment of Grooved Pegboard Test, 25 Pegs Group at Week 12: Active Comparator Phase/Efficacy Phase
Description: The grooved pegboard test was a manipulative dexterity test that assessed psychomotor speed, fine motor control, and rapid-visual motor coordination. It consisted of a small board of 25 holes with randomly positioned slots. Pegs with a key along one side must be rotated to match the hole before they can be inserted. Participants were asked to insert 25 grooved pegs into the holes within the given time limit (up to 300 seconds). In this outcome measure number of pegs dropped while putting in the holes were measured. The task needs to be completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand.
Time Frame: Baseline, Week 12
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: pegs
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 33 | 34 | 33 | 10 | 9
pegs
  Dominant hand: Baseline | 0.45 (1.20) | 0.24 (0.50) | 0.24 (0.66) | 0.10 (0.32) | 0.11 (0.33)
  Dominant hand: Change at Week 12: number analyzed (Participants) | 30 | 33 | 33 | 8 | 9
  Dominant hand: Change at Week 12 | 0.00 (1.05) | -0.18 (0.58) | 0.09 (0.77) | 0.00 (0.53) | 0.44 (1.33)
  Non-dominant hand: Baseline: number analyzed (Participants) | 33 | 32 | 33 | 10 | 8
  Non-dominant hand: Baseline | 0.91 (2.36) | 0.28 (0.46) | 0.36 (0.78) | 0.40 (0.97) | 0.13 (0.35)
  Non-dominant hand: Change at Week 12: number analyzed (Participants) | 30 | 31 | 33 | 8 | 8
  Non-dominant hand: Change at Week 12 | -0.33 (1.60) | 0.06 (1.03) | 0.21 (1.78) | 0.13 (0.35) | 0.00 (0.00)

31. Secondary Outcome: Change From Baseline in Number of Pegs Dropped Assessment of Grooved Pegboard Test, 25 Pegs Group at Week 24: Safety Extension Phase
Description: as for outcome 30
Time Frame: Baseline, Week 24
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: pegs
Arm/Group | Cohort 1, Safety Extension Phase: Fesoterodine 4 mg | Cohort 1, Safety Extension Phase: Fesoterodine 8 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg Then 8 mg | Cohort 2, Safety Extension Phase: Fesoterodine 2 mg | Cohort 2, Safety Extension Phase: Fesoterodine 4 mg
Number analyzed (Participants) | 25 | 30 | 14 | 16 | 5 | 9
pegs
  Dominant hand: Change at Week 24 | 0.00 (0.87) | 0.63 (4.63) | 0.14 (0.36) | 0.25 (1.24) | 0.00 (0.00) | 0.44 (1.33)
  Non-dominant hand: Change at Week 24: number analyzed (Participants) | 25 | 28 | 14 | 15 | 5 | 8
  Non-dominant hand: Change at Week 24 | -0.28 (2.17) | 0.68 (4.79) | 0.00 (0.39) | 0.27 (1.67) | 0.60 (0.89) | -0.13 (0.35)

32. Secondary Outcome: Change From Baseline in Number of Pegs Placed Correctly Assessment of Grooved Pegboard Test, 10 Pegs Group at Week 12: Active Comparator Phase/Efficacy Phase
Description: The grooved pegboard test was a manipulative dexterity test that assessed psychomotor speed, fine motor control, and rapid-visual motor coordination. It consisted of a small board of 25 holes with randomly positioned slots. Pegs with a key along one side must be rotated to match the hole before they can be inserted. Participants were asked to insert 10 grooved pegs into the holes within the given time limit (up to 300 seconds). In this outcome measure number of pegs placed correctly while putting in the holes were measured. The task needs to be completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand.
Time Frame: Baseline, Week 12
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: pegs
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 9 | 9 | 7 | 18 | 21
pegs
  Dominant hand: Baseline: number analyzed (Participants) | 9 | 8 | 7 | 18 | 20
  Dominant hand: Baseline | 9.56 (1.01) | 9.38 (1.77) | 10.00 (0.00) | 9.89 (0.47) | 10.0 (0.00)
  Dominant hand: Change at Week 12: number analyzed (Participants) | 7 | 7 | 6 | 15 | 19
  Dominant hand: Change at Week 12 | -0.29 (0.76) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.38) | -0.11 (0.46)
  Non-dominant hand: Baseline: number analyzed (Participants) | 9 | 9 | 7 | 17 | 21
  Non-dominant hand: Baseline | 9.56 (1.01) | 9.00 (2.35) | 10.00 (0.00) | 9.82 (0.73) | 9.62 (1.20)
  Non-dominant hand: Change at Week 12: number analyzed (Participants) | 7 | 6 | 6 | 14 | 20
  Non-dominant hand: Change at Week 12 | -0.57 (1.13) | 0.00 (0.00) | 0.00 (0.00) | -0.07 (0.62) | 0.00 (0.32)

33. Secondary Outcome: Change From Baseline in Number of Pegs Placed Correctly Assessment of Grooved Pegboard Test, 10 Pegs Group at Week 24: Safety Extension Phase
Description: as for outcome 32
Time Frame: Baseline, Week 24
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: pegs
Arm/Group | Cohort 1, Safety Extension Phase: Fesoterodine 4 mg | Cohort 1, Safety Extension Phase: Fesoterodine 8 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg Then 8 mg | Cohort 2, Safety Extension Phase: Fesoterodine 2 mg | Cohort 2, Safety Extension Phase: Fesoterodine 4 mg
Number analyzed (Participants) | 3 | 7 | 2 | 3 | 15 | 19
pegs
  Dominant hand: Change at Week 24: number analyzed (Participants) | 3 | 7 | 2 | 3 | 15 | 18
  Dominant hand: Change at Week 24 | -0.33 (0.58) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.07 (0.26) | 0.00 (0.00)
  Non-dominant hand: Change at Week 24: number analyzed (Participants) | 3 | 6 | 2 | 3 | 14 | 19
  Non-dominant hand: Change at Week 24 | -1.33 (2.31) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.14 (0.53) | 0.21 (0.92)

34. Secondary Outcome: Change From Baseline in Number of Pegs Placed Correctly Assessment of Grooved Pegboard Test, 25 Pegs Group at Week 12: Active Comparator Phase/Efficacy Phase
Description: The grooved pegboard test was a manipulative dexterity test that assessed psychomotor speed, fine motor control, and rapid-visual motor coordination. It consisted of a small board of 25 holes with randomly positioned slots. Pegs with a key along one side must be rotated to match the hole before they can be inserted. Participants were asked to insert 25 grooved pegs into the holes within the given time limit (up to 300 seconds). In this outcome measure number of pegs placed correctly while putting in the holes were measured. The task needs to be completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand.
Time Frame: Baseline, Week 12
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: pegs
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 33 | 34 | 33 | 10 | 9
pegs
  Dominant hand: Baseline | 25.00 (0.00) | 24.56 (1.89) | 25.00 (0.00) | 25.00 (0.00) | 23.22 (3.83)
  Dominant hand: Change at Week 12: number analyzed (Participants) | 30 | 33 | 33 | 8 | 9
  Dominant hand: Change at Week 12 | -0.07 (0.25) | 0.42 (1.77) | -0.12 (0.70) | -0.13 (0.35) | 0.11 (2.76)
  Non-dominant hand: Baseline: number analyzed (Participants) | 33 | 32 | 33 | 10 | 8
  Non-dominant hand: Baseline | 24.45 (2.09) | 24.75 (0.92) | 24.88 (0.42) | 24.50 (1.58) | 24.25 (1.75)
  Non-dominant hand: Change at Week 12: number analyzed (Participants) | 30 | 31 | 33 | 8 | 8
  Non-dominant hand: Change at Week 12 | 0.53 (2.19) | 0.26 (0.93) | 0.03 (0.30) | 0.63 (1.77) | -0.63 (1.77)

35. Secondary Outcome: Change From Baseline in Number of Pegs Placed Correctly Assessment of Grooved Pegboard Test, 25 Pegs Group at Week 24: Safety Extension Phase
Description: as for outcome 34
Time Frame: Baseline, Week 24
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: pegs
Arm/Group | Cohort 1, Safety Extension Phase: Fesoterodine 4 mg | Cohort 1, Safety Extension Phase: Fesoterodine 8 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg Then 8 mg | Cohort 2, Safety Extension Phase: Fesoterodine 2 mg | Cohort 2, Safety Extension Phase: Fesoterodine 4 mg
Number analyzed (Participants) | 25 | 30 | 14 | 16 | 5 | 9
pegs
  Dominant hand: Change at Week 24 | 0.00 (0.00) | 0.50 (2.01) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.11 (2.76)
  Non-dominant hand: Change at Week 24: number analyzed (Participants) | 25 | 28 | 14 | 15 | 5 | 8
  Non-dominant hand: Change at Week 24 | 0.60 (2.40) | 0.21 (0.96) | 0.14 (0.66) | 0.00 (0.00) | 0.60 (2.61) | -0.50 (1.85)

36. Secondary Outcome: Number of Participants Meeting Pre-defined Criteria for Vital Signs Values From Baseline Through Week 12: Active Comparator/Efficacy Phase
Description: Pre-defined criteria for vital signs: 1) a) systolic blood pressure (SBP) of <90 millimeter of mercury (mmHg), b) change >=30 mmHg increase, c) change >=30 mmHg decrease; 2) a) diastolic blood pressure (DBP) of <50 mmHg, b) change >=20 mmHg increase, c) change >=20 mmHg decrease; 3) a) pulse rate value of <40 beats per minute (bpm), b) pulse rate value >120 bpm.
Time Frame: Baseline up to Week 12
Population: Analysis set population for active comparator phase and efficacy phase: all participants of respective cohorts who received at least 1 dose of study medication in relevant phase. Here, "Overall Number of Participants Analyzed": participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 40 | 41 | 40 | 24 | 29
Participants
  SBP: <90 mmHg | 2 | 2 | 0 | 7 | 4
  SBP: Change >=30 mmHg increase | 1 | 2 | 1 | 0 | 1
  SBP: Change >=30 mmHg decrease | 1 | 0 | 0 | 0 | 0
  DBP: <50 mmHg | 2 | 1 | 2 | 3 | 1
  DBP: Change >=20 mmHg increase | 1 | 2 | 1 | 3 | 4
  DBP: Change >=20 mmHg decrease | 1 | 1 | 1 | 2 | 0
  Pulse rate: <40 bpm | 0 | 0 | 0 | 0 | 0
  Pulse rate: >120 bpm | 2 | 4 | 0 | 2 | 3

37. Secondary Outcome: Number of Participants Meeting Pre-defined Criteria for Vital Signs Values From Baseline Through Week 24: Safety Extension Phase
Description: as for outcome 36
Time Frame: Baseline up to Week 24
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Safety Extension Phase: Fesoterodine 4 mg | Cohort 1, Safety Extension Phase: Fesoterodine 8 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg Then 8 mg | Cohort 2, Safety Extension Phase: Fesoterodine 2 mg | Cohort 2, Safety Extension Phase: Fesoterodine 4 mg
Number analyzed (Participants) | 30 | 37 | 16 | 20 | 20 | 28
Participants
  SBP: <90 mmHg | 0 | 3 | 2 | 1 | 4 | 2
  SBP: Change >=30 mmHg increase | 1 | 0 | 0 | 0 | 0 | 0
  SBP: Change >=30 mmHg decrease | 0 | 1 | 0 | 0 | 0 | 0
  DBP: <50 mmHg | 0 | 2 | 0 | 0 | 2 | 0
  DBP: Change >=20 mmHg increase | 1 | 0 | 0 | 0 | 1 | 2
  DBP: Change >=20 mmHg decrease | 1 | 0 | 0 | 0 | 0 | 0
  Pulse rate: <40 bpm | 0 | 0 | 0 | 0 | 0 | 0
  Pulse rate: >120 bpm | 0 | 0 | 0 | 0 | 0 | 1

38. Secondary Outcome: Number of Participants With Clinically Significant Urinary Tract Infections (UTI): Active Comparator/Efficacy Phase
Description: Clinically significant UTI, counted as an adverse event was defined as: positive urine culture with a uropathogen (defined as >=10^5 colony forming unit per milliliter [CFU/mL]) and the presence of symptoms, or pyuria (defined as >50 white blood cells [WBC] per high-pass filter [hpf]) and the presence of symptoms, or positive urine culture with a uropathogen (defined as >=10^5 CFU/mL) with or without symptoms in a participant with a documented history of vesicoureteral reflux (VUR).
Time Frame: Week 1 up to Week 12
Population: Safety analysis set population for active comparator phase and efficacy phase: all participants of respective cohorts who received at least 1 dose of study medication in relevant phase of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 42 | 42 | 40 | 28 | 29
Participants | 4 | 1 | 4 | 3 | 4

39. Secondary Outcome: Number of Participants With Clinically Significant Urinary Tract Infections (UTI): Safety Extension Phase
Description: Clinically significant UTI, counted as an adverse event was defined as: positive urine culture with a uropathogen (defined as >=10^5 CFU/mL) and the presence of symptoms, or pyuria (defined as >50 WBC per hpf and the presence of symptoms, or positive urine culture with a uropathogen (defined as >=10^5 CFU/mL) with or without symptoms in a participants with a documented history of VUR.
Time Frame: Week 12 up to Week 26
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Safety Extension Phase: Fesoterodine 4 mg | Cohort 1, Safety Extension Phase: Fesoterodine 8 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg Then 8 mg | Cohort 2, Safety Extension Phase: Fesoterodine 2 mg | Cohort 2, Safety Extension Phase: Fesoterodine 4 mg
Number analyzed (Participants) | 30 | 37 | 16 | 20 | 20 | 28
Participants | 0 | 1 | 2 | 0 | 1 | 5

40. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities: Active Comparator/Efficacy Phase
Description: Hematology: hemoglobin, hematocrit, erythrocytes <0.8*lower limit of normal (LLN), platelets<0.5*LLN>1.75*upper limit of normal (ULN), leukocytes <0.6*LLN>1.5*ULN, lymphocytes, neutrophils, <0.8*LLN >1.2*ULN, basophils, eosinophils, monocytes monocytes/leukocytes >1.2*ULN. Clinical chemistry: bilirubin, direct, bilirubin >1.5*ULN, aspartate aminotransferase (AT), alanine AT, gamma glutamyl transferase, lactate dehydrogenase, alkaline phosphatase>3.0*ULN, protein, albumin, phosphate <0.8*LLN >1.2*ULN, blood urea nitrogen, creatinine >1.3*ULN, urate >1.2*ULN, sodium<0.95*LLN>1.05*ULN, potassium, chloride, calcium bicarbonate<0.9*LLN>1.1*ULN, glucose<0.6*LLN>1.5*ULN, creatine kinase >2.0*ULN. Urinalysis: specific gravity <1.003>1.030, pH <4.5>8, urine glucose, ketones, urine protein, urine hemoglobin, urine bilirubin, nitrite, >=1, urine erythrocytes, urine leukocytes >=20, epithelial cells >=6, bacteria >20.
Time Frame: Week 1 up to Week 12
Population: Safety analysis set population for active comparator phase and efficacy phase: all participants of respective cohorts who received at least 1 dose of study medication in relevant phase. Here, "Overall Number of Participants Analyzed": participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 39 | 41 | 39 | 24 | 29
Participants | 30 | 29 | 27 | 19 | 19

41. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities: Safety Extension Phase
Description: as for outcome 40
Time Frame: Week 12 up to Week 26
Population: Safety analysis set population for safety extension phase: all participants of respective cohorts who received at least 1 dose of study medication in the relevant phase. Here, "Overall Number of Participants Analyzed": participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Safety Extension Phase: Fesoterodine 4 mg | Cohort 1, Safety Extension Phase: Fesoterodine 8 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg Then 8 mg | Cohort 2, Safety Extension Phase: Fesoterodine 2 mg | Cohort 2, Safety Extension Phase: Fesoterodine 4 mg
Number analyzed (Participants) | 30 | 36 | 16 | 19 | 20 | 28
Participants | 19 | 22 | 7 | 12 | 15 | 21

42. Secondary Outcome: Change From Baseline in Post-Void Residual (PVR) Volume at Weeks 4, 12: Active Comparator Phase/Efficacy Phase
Description: Post-void residual volume measurement was measured by an ultrasound. PVR volume was only assessed for participants who did not perform clean intermittent catheterization or in any participants who had >1 UTI during the study.
Time Frame: Baseline, Week 4, 12
Population: Safety analysis set population for active comparator phase and efficacy phase: all participants of respective cohorts who received at least 1 dose of study medication in relevant phase. Here, "Overall Number of Participants Analyzed": participants evaluable for this outcome measure; "Number Analyzed": participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 6 | 7 | 9 | 6 | 6
milliliter
  Baseline | 7.00 (8.20) | 9.57 (12.54) | 5.78 (7.98) | 14.7 (14.31) | 10.7 (7.94)
  Change at Week 4: number analyzed (Participants) | 5 | 6 | 9 | 3 | 4
  Change at Week 4 | 5.40 (7.60) | -7.33 (10.88) | 19.11 (24.52) | -2.00 (6.24) | 10.25 (34.40)
  Change at Week 12: number analyzed (Participants) | 5 | 6 | 7 | 4 | 4
  Change at Week 12 | 25.60 (53.42) | -4.00 (8.41) | 12.86 (43.48) | 2.50 (16.05) | 0.75 (17.46)

43. Secondary Outcome: Change From Baseline in Post-Void Residual Volume at Week 24: Safety Extension Phase
Description: as for outcome 42
Time Frame: Baseline, Week 24
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Cohort 1, Safety Extension Phase: Fesoterodine 4 mg | Cohort 1, Safety Extension Phase: Fesoterodine 8 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg Then 8 mg | Cohort 2, Safety Extension Phase: Fesoterodine 2 mg | Cohort 2, Safety Extension Phase: Fesoterodine 4 mg
Number analyzed (Participants) | 4 | 5 | 5 | 3 | 3 | 4
milliliter | 11.50 (23.67) | 11.60 (29.43) | 18.00 (31.36) | 36.67 (59.23) | 21.67 (20.21) | 2.75 (14.50)

44. Secondary Outcome: Number of Participants With Clinically Relevant Changes in Physical Examination Findings From Baseline to Week 12: Active Comparator/Efficacy Phase
Description: Physical examination included assessment of the general appearance and the skin, head, ears, eyes, nose, mouth, throat, respiratory, cardiovascular, gastrointestinal, musculoskeletal and neurological systems. Clinically relevant changes in physical findings were assessed by the investigator.
Time Frame: Baseline up to Week 12
Population: Safety analysis set population for active comparator phase and efficacy phase: all participants of respective cohorts who received at least 1 dose of study medication in relevant phase of the study. Here, "Overall Number of Participants Analyzed": participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg Then 4 mg
Number analyzed (Participants) | 38 | 42 | 40 | 28 | 29
Participants | 2 | 1 | 1 | 1 | 0

45. Secondary Outcome: Number of Participants With Clinically Relevant Changes in Physical Examination Findings From Baseline to Week 24: Safety Extension Phase
Description: as for outcome 44
Time Frame: Baseline up to Week 24
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Safety Extension Phase: Fesoterodine 4 mg | Cohort 1, Safety Extension Phase: Fesoterodine 8 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg Then 8 mg | Cohort 2, Safety Extension Phase: Fesoterodine 2 mg | Cohort 2, Safety Extension Phase: Fesoterodine 4 mg
Number analyzed (Participants) | 30 | 37 | 16 | 20 | 20 | 28
Participants | 3 | 2 | 0 | 0 | 0 | 2

46. Secondary Outcome: Absorption Rate Constant (Ka) of Fesoterodine
Description: Absorption rate constant is used to determine rate at which drug is entering into body. Pharmacokinetic (PK) analysis was not done separately for each dose of fesoterodine in respective cohorts and were combined for PK analysis using PK modelling approach.
Time Frame: Week 4, Day 1: pre-dose (when dose administered at clinic) or if dose taken at home up to 3 hours before coming to the clinic, sampling just after arrival at clinic, 5 hours post-dose, 8-10 hours post-dose (if participants remained at clinic)
Population: The PK analysis population included all participants randomized and treated with fesoterodine and who had at least 1 of the PK parameters of primary interest during the study.
Measure: Mean (Standard Error); unit: per hour
Groups:
- Fesoterodine Pooled: Participants received any dose of fesoterodine in the study from Week 1 to Week 24.
Arm/Group | Fesoterodine Pooled
Number analyzed (Participants) | 121
per hour | 0.0897 (5.99)

47. Secondary Outcome: Apparent Oral Clearance (CL/F) of Fesoterodine
Description: Clearance determines the rate at which a drug is metabolized or eliminated by normal biological processes. PK analysis was not done separately for each dose of fesoterodine in respective cohorts and were combined for PK analysis using PK modelling approach.
Time Frame: as for outcome 46
Population: as for outcome 46
Measure: Mean (Standard Error); unit: liter per hour
Arm/Group | Fesoterodine Pooled
Number analyzed (Participants) | 121
liter per hour | 71.6 (6.7)

48. Secondary Outcome: Volume of Distribution (Vd) of Fesoterodine
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. PK analysis was not done separately for each dose of fesoterodine in respective cohorts and were combined for PK analysis using PK modelling approach.
Time Frame: as for outcome 46
Population: as for outcome 46
Measure: Mean (Standard Error); unit: liter
Arm/Group | Fesoterodine Pooled
Number analyzed (Participants) | 121
liter | 68.1 (29.7)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 26 (includes 2 week of follow up)
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis population evaluated.
Groups:
- Cohort 1,SEP: Oxybutynin Then Fesoterodine 8 mg: Participants with body weight >25 kg who were randomized to receive oxybutynin ER tablet, at a daily dose in accordance with approved pediatric labeling and accepted practice, in active comparator phase; were allocated by investigator to receive fesoterodine 4 mg PR tablet orally once daily for first 1 week followed by fesoterodine 8 mg PR tablet orally once daily for another 11 weeks (if the fesoterodine 4 mg dose was well tolerated) in the safety extension phase and if dose was not tolerated participants were withdrawn from the study.
- Cohort 2 Efficacy Phase: Fesoterodine 4 mg: Participants with body weight <=25 kg were randomized to receive fesoterodine 2 mg BIC capsule orally once daily for first 1 week and if dose was tolerated well, participants received 4 mg BIC capsule orally once daily for next 11 weeks in efficacy phase and if dose was not tolerated then participants were withdrawn from the study.
Arm/Group | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg | Cohort 1, Active Comparator Phase: Oxybutynin | Cohort 1, Safety Extension Phase: Fesoterodine 4 mg | Cohort 1, Safety Extension Phase (SEP): Fesoterodine 8 mg | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg | Cohort 1,SEP: Oxybutynin Then Fesoterodine 8 mg | Cohort 2, Efficacy Phase: Fesoterodine 2 mg | Cohort 2 Efficacy Phase: Fesoterodine 4 mg | Cohort 2, Safety Extension Phase: Fesoterodine 2 mg | Cohort 2, Safety Extension Phase: Fesoterodine 4 mg
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42 | 0/40 | 0/30 | 0/37 | 0/16 | 0/20 | 0/28 | 0/29 | 0/20 | 0/28
Serious Adverse Events (participants affected / at risk) | 3/42 | 2/42 | 1/40 | 0/30 | 2/37 | 0/16 | 0/20 | 2/28 | 2/29 | 0/20 | 2/28
Other Adverse Events (participants affected / at risk) | 26/42 | 19/42 | 30/40 | 14/30 | 13/37 | 9/16 | 11/20 | 19/28 | 17/29 | 11/20 | 14/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg (N=42) | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg (N=42) | Cohort 1, Active Comparator Phase: Oxybutynin (N=40) | Cohort 1, Safety Extension Phase: Fesoterodine 4 mg (N=30) | Cohort 1, Safety Extension Phase (SEP): Fesoterodine 8 mg (N=37) | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg (N=16) | Cohort 1,SEP: Oxybutynin Then Fesoterodine 8 mg (N=20) | Cohort 2, Efficacy Phase: Fesoterodine 2 mg (N=28) | Cohort 2 Efficacy Phase: Fesoterodine 4 mg (N=29) | Cohort 2, Safety Extension Phase: Fesoterodine 2 mg (N=20) | Cohort 2, Safety Extension Phase: Fesoterodine 4 mg (N=28)
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Complicated appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg (N=42) | Cohort 1, Active Comparator Phase: Fesoterodine 4 mg Then 8 mg (N=42) | Cohort 1, Active Comparator Phase: Oxybutynin (N=40) | Cohort 1, Safety Extension Phase: Fesoterodine 4 mg (N=30) | Cohort 1, Safety Extension Phase (SEP): Fesoterodine 8 mg (N=37) | Cohort 1, SEP: Oxybutynin Then Fesoterodine 4 mg (N=16) | Cohort 1,SEP: Oxybutynin Then Fesoterodine 8 mg (N=20) | Cohort 2, Efficacy Phase: Fesoterodine 2 mg (N=28) | Cohort 2 Efficacy Phase: Fesoterodine 4 mg (N=29) | Cohort 2, Safety Extension Phase: Fesoterodine 2 mg (N=20) | Cohort 2, Safety Extension Phase: Fesoterodine 4 mg (N=28)
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Astigmatism (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myopia (Eye disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Strabismus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 3 | 5 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 3 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 4 | 11 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 1 | 1 | 1 | 1 | 2 | 0 | 1 | 2 | 2 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 2 | 3 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infection parasitic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 4 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mastitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 5 | 1 | 2 | 1 | 2 | 1 | 2 | 3 | 3 | 2 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 2
Urinary tract infection (Infections and infestations) | 3 | 1 | 3 | 0 | 1 | 2 | 0 | 2 | 3 | 1 | 4
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacterial test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Investigation abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Residual urine volume increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urine analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 5 | 1 | 3 | 1 | 1 | 0 | 2 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Behaviour disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Incontinence (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Genital pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheelchair user (Social circumstances) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis infected (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear lobe infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Accommodation disorder (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip erythema (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adverse drug reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thirst (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine output increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encopresis (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urethral pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine flow decreased (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystogram (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2014-03-03): https://cdn.clinicaltrials.gov/large-docs/44/NCT01557244/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT01557244/SAP_001.pdf